Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

# STATISTICAL ANALYSIS PLAN

# Medivir AB

### Protocol MIV-711-201

A Randomised, Double-blind Placebo-controlled Phase IIa Study to Evaluate Efficacy, Safety and Tolerability of MIV-711 in Knee Joint Osteoarthritis

PAREXEL Study Number: 226198

Version: Final 1.0 Date: 22 June 2017

Medivir Protocol: MIV-711-201 Final 1.0 22 June 2017

# SIGNATURE PAGE - MEDIVIR

# **Declaration**

The undersigned agree to the statistical analyses and procedures of this clinical study.

| John Old | 22-JUN-2017 |
|---|---|
| John Öhd<br>MD PhD<br>Director Clinical R&D<br>Medivir AB | Date (dd mmm yyyy) |

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

# **SIGNATURE PAGE - PAREXEL**

# **Delaration**

The undersigned agree to the statistical analyses and procedures of this clinical study.

Date (dd mmm yyyy)

Prepared by:

Walter Heber, MSc

Associate Manager, EP Biostatistics PAREXEL International Corporation

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

# **TABLE OF CONTENTS**

| SIGNA | ATURE PAGE - MEDIVIR | 2 |
|-------|--------------------------------------|----|
| SIGNA | ATURE PAGE - PAREXEL | 3 |
| TABL | E OF CONTENTS | 4 |
| 1. | STATISTICAL ANALYSIS PLAN | 9 |
| 2. | STUDY OBJECTIVES AND HYPOTHESES | 9 |
| 2.1.1 | PRIMARY OBJECTIVE | 9 |
| 2.1.2 | HYPOTHESIS TO BE TESTED. | 9 |
| 2.2 | SECONDARY OBJECTIVES | 9 |
| 2.3 | EXPLORATORY OBJECTIVES | 10 |
| 2.3.1 | BIOMARKERS | 10 |
| 2.3.2 | PHARMACOKINETICS | 10 |
| 3. | STUDY DESIGN | 11 |
| 3.1 | STUDY ENDPOINTS | 11 |
| 3.1.1 | PRIMARY ENDPOINT | 11 |
| 3.1.2 | SECONDARY ENDPOINT | 12 |
| 3.1.3 | OTHER SECONDARY ENDPOINTS | 12 |
| 3.1.4 | SAFETY ENDPOINTS | 12 |
| 3.2 | STUDY POPULATION | 13 |
| 3.3 | SAMPLE SIZE ESTIMATION | 13 |
| 3.4 | DOSE ADMINISTRATION | 13 |
| 3.5 | RANDOMIZATION | 14 |
| 3.6 | PATIENT REPLACEMENT | 14 |
| 3.7 | TRIAL BLINDING | 14 |
| 3.8 | PROTOCOL DEVIATIONS | 14 |
| 3.9 | INTERIM ANALYSIS | 15 |
| 3.10 | EXTENSION PROTOCOL | 15 |
| 4. | STUDY ANALYSIS VARIABLES | 15 |
| 4.1 | DEMOGRAPHIC AND BACKGROUND VARIABLES | 15 |
| 4.2 | SAFETY VARIABLES | 16 |
| 4.2.1 | ADVERSE EVENTS | 16 |
| 4.2.2 | CLINICAL LABORATORY TESTS | 16 |

| Medivir<br>Protocol: | Fina 22 June 2 | |
|---|---|---|
| 4.2.3 | OTHER LABORATORY TESTS | 16 |
| 4.2.4 | VITAL SIGNS | 17 |
| 4.2.5 | ELECTROCARDIOGRAMS | 17 |
| 4.2.6 | PHYSICAL EXAMINATION | 17 |
| 4.2.7 | PRIOR AND CONCOMITANT MEDICATIONS | 17 |
| 4.2.8 | ADHERENCE TO STUDY MEDICATIONS | 18 |
| 4.2.9 | PHONE CALL TO ASSESS SAFETY AND TOLERABILITY | 18 |
| 4.3 | PHARMACODYNAMIC VARIABLES - EFFICACY | 18 |
| 4.3.1 | PAIN | 18 |
| 4.3.2 | MRI AND IMAGING | 18 |
| 4.3.3 | PATIENT REPORTED OUTCOMES (PRO) | 20 |
| 4.3.3.1 | NRS SCORES - KNEE PAIN AND FUNCTION IN THE LAST WEEK | 20 |
| 4.3.3.2 | ICOAP SCORES | 21 |
| 4.3.3.3 | WOMAC SCORES | 21 |
| 4.3.3.4 | OMERACT SCORES | 22 |
| 4.3.3.5 | GLOBAL IMPROVEMENT SCORES | 22 |
| 4.3.3.6 | QUALITY OF LIFE | 23 |
| 4.3.3.7 | BRIEF MEDICATION QUESTIONNAIRE | 23 |
| 4.3.3.8 | E-DIARY ASSESSNMENT OF NRS AND ANALGESIC USE | 23 |
| 4.3.4 | SECONDARY EFFICACY PARAMETERS | 24 |
| 4.3.4.1 | BIOMARKERS | 24 |
| 4.3.4.2 | OTHER IMAGING ASSESSMENTS | 24 |
| 4.4 | ANALYSIS POPULATIONS | 24 |
| 4.4.1 | INTENT-TO-TREAT POPULATION (ITT) | 24 |
| 4.4.2 | MODIFIED INTENT-TO-TREAT POPULATION (MITT) | |
| 4.4.3 | PER PROTOCOL POPULATION (PPS) | |
| 4.4.4 | SAFETY ANALYSIS POPULATION (SAF) | 25 |
| 5. | GENERAL CONSIDERATIONS FOR DATA PRESENTATIONS | 25 |
| 5.1 | SOFTWARE | 26 |
| 6. | PATIENT AND TREATMENT INFORMATION | 26 |
| 6.1 | PATIENT DISPOSITION | 26 |
| 6.2 | PATIENTS EXCLUDED FROM ANALYSIS POPULATIONS | 27 |
| 6.3 | ELIGIBILITY CRITERIA | 27 |

| Medivir<br>Protocol: | MIV-711-201 22 | Final 1.0<br>June 2017 |
|---|---|---|
| 6.4 | EXCLUSION TESTS | 27 |
| 6.5 | PROTOCOL DEVIATIONS | 27 |
| 6.6 | DEMOGRAPHIC DATA | 27 |
| 6.7 | MEDICAL HISTORY | 27 |
| 6.8 | PRIOR AND CONCOMITANT MEDICATION | 28 |
| 6.9 | DOSE ADMINISTRATION | 28 |
| 7. | PHARMACODYNAMIC ANALYSIS - EFFICACY | 28 |
| 7.1 | NRS PAIN DATA | 28 |
| 7.2 | STATISTICAL ANALYSIS OF THE NRS PAIN DATA | 29 |
| 7.2.1 | MULTIPLICITY ADJUSTMENT FOR THE PRIMARY ENDPOINT | 31 |
| 7.2.2 | VISUALIZATIONS FOR THE PRIMARY ENDPOINT | 31 |
| 7.3 | KEY SECONDARY ANALYSIS: MRI OF BONE AREA IN TARC | |
| 7.3.1 | STATISTICAL ANALYSIS OF THE MRI OF BONE AREA IN TARCKNEE | _ |
| 7.4 | SECONDARY ANALYSIS: MRI OF CARTILAGE THICKNESS TARGET KNEE | |
| 7.4.1 | STATISTICAL ANALYSIS OF THE MRI OF CARTILAGE THICKN IN TARGET KNEE. | |
| 7.5 | SECONDARY ANALYSIS: MRI OF TOTAL BML VOLUME TARGET KNEE | IN |
| 7.5.1 | STATISTICAL ANALYSIS OF THE MRI OF TOTAL BML VOLUME TARGET KNEE | E IN |
| 7.6 | ANALYSIS OF OTHER SECONDARY IMAGING ASSESSMENTS | 33 |
| 7.7 | ANALYSIS OF OTHER PATIENT REPORTED OUTCOMES (PROS). | 34 |
| 7.7.1 | INTERMITTENT AND CONSTANT OSTEOARTHRITIS PAIN (ICO KNEE VERSION | |
| 7.7.2 | ANALYSIS OF THE WOMAC | 35 |
| 7.7.3 | (OARSI)-OMERACT RESPONDER CRITERIA | 35 |
| 7.7.4 | GLOBAL IMPROVEMENTS | |
| 7.7.5 | QUALITY OF LIFE PRO – EQ-5D-5L | 37 |
| 7.7.6 | E-DIARY FOR PATIENT PAIN | 38 |
| 7.7.7 | BIOMARKERS FROM SERUM AND URINE SAMPLES | 38 |
| 8. | SAFETY ANALYSIS | 39 |
| 8.1 | ADVERSE EVENTS | 39 |

| Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017 | | |
|---|---|---|
| 8.2 | CLINICAL SAFETY LABORATORY TESTS (HEMATOLOGY, CHEMISTRY, URINALYSIS) | 40 |
| 8.2.1 | HEMATOLOGY AND CHEMISTRY | 40 |
| 8.2.2 | URINALYSIS | 41 |
| 8.3 | OTHER BLOOD AND URINE SAMPLES | 41 |
| 8.4 | VITAL SIGNS | 41 |
| 8.5 | 12-LEAD SAFETY ECG | 41 |
| 8.6 | PHYSICAL EXAMINATION AND WEIGHT | 42 |
| 8.7 | PHONE CALL TO ASSESS SAFETY | 42 |
| 9. | REPORTING OUTPUT | 43 |
| 10. | REFERENCES | 44 |
| 11. | SUMMARY TABLES | 45 |
| 12. | FIGURES | 48 |
| 13. | LISTINGS | 50 |
| 14. | TABLE SHELLS | 52 |
| 15. | LISTING SHELLS | 103 |

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

### Abbreviations and definitions

AE Adverse event

BLQ Below the lower limit of quantification

BMI Body Mass Index
BML Bone Marrow Lesions
CI Confidence interval
CS Clinically significant
CV Coefficient of variation
ECG Electrocardiogram
FAS Full analysis set

h Hour

HBsAg Hepatitis B surface antigen

HCV Hepatitis C virus

HIV Human immunodeficiency virus
IMP Investigational Medicinal Product
LLOQ Lower limit of quantification

MedDRA Medical Dictionary for Regulatory Activities

MOAKS MRI Osteoarthritis Knee Score NCS Not clinically significant NRS Numeric Rating Scale

NK Not known
OA Osteoarthritis
PK Pharmacokinetic
OOL Quality of Life

SAE Serious adverse event
SAP Statistical Analysis Plan
SD Standard deviation
SOC System Organ Class

t½ Apparent terminal elimination half-life
TEAE Treatment-emergent adverse event
TIC Time Integrated Concentrations

Tmax Time corresponding to occurrence of Cmax WHO-DD World Health Organisation - Drug Dictionary

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

# 1. Statistical Analysis Plan

This Statistical Analysis Plan (SAP) is based on the final protocol, dated 09 September 2015 as well as all protocol amendments finalized including: amendment 1 dated 13 January 2016 and amendment 2 dated 20 July 2016. The SAP provides details on the planned statistical methodology for the primary and secondary analysis of the study data. The SAP also outlines the statistical programming specifications for the tables, listings and figures. It describes the safety and pharmacodynamic (PD) data, the handling of that data; the anticipated data transformations and manipulations, and other details of the analyses not provided in the study protocol. This SAP covers the planned analysis to be conducted by PAREXEL of all safety and efficacy data as described in the protocol, and as collected in the source data.

# 2. Study Objectives and Hypotheses

### 2.1.1 Primary Objective

To assess the effect of MIV-711 on knee pain (at week 26), as measured by an 11-point numerical rating scale in patients with symptomatic and radiographic knee osteoarthritis

### 2.1.2 Hypothesis to be Tested

The primary hypothesis of this study is that MIV-711 will reduce pain in patients with moderate knee osteoarthritis diagnosed based on symptomatic and radiologic criteria.

## 2.2 Secondary Objectives

To assess the effect of MIV-711 on MRI target knee bone area in patients with symptomatic and radiographic knee OA over 26 weeks.

Other secondary objectives include:

To assess, in patients with symptomatic and radiographic knee OA, over 26 weeks:

- \*The effect of MIV-711 on worst target knee pain (1 week recall)
- The effect of MIV-711 on average contralateral knee pain (1 week recall)
- \*The effect of MIV-711 on constant and intermittent OA pain
- \*The effect of MIV-711 on global improvements in knee problem, knee pain and knee function
- \*The effect of MIV-711 on knee joint OA symptoms (function, pain, stiffness)
- The effect of MIV-711 on global disease activity
- The effect of MIV-711 on quality of life (QOL)

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

- \*The effect of MIV-711 on MRI bone area in regions other than primary region
- \*The effect of MIV-711 on MRI bone marrow lesion volume
- \*The effect of MIV-711 on MRI cartilage thickness loss
- The effect of MIV-711 in the semi quantitative MRI Osteoarthritis Knee Score (MOAKS) parameters
- \*The effect of MIV-711 on patient reported e-diary daily recall knee joint pain
- The effect of MIV-711 on patient reported e-diary daily recall analgesics use
- The safety and tolerability of MIV-711
- The effect of MIV-711 on biomarkers for bone resorption (serum CTX-I) and for cartilage degradation (urine CTX-II) assessment

### 2.3 Exploratory Objectives

In addition, the study will address the following exploratory objectives.

#### 2.3.1 Biomarkers

- Assessment of the effect of MIV-711 on serum and urinary biomarkers of relevance for OA
- Serum CTXI and urine CTXII will be the only biomarkers covered in this SAP; all other biomarkers mentioned in the study protocol will not be included in this SAP.
- Baseline (visit 2) and steady state treatment (visit 8) blood and urinary samples will be stored for patients who sign a separate voluntary Informed Consent Form (ICF) for potential future pharmacogenomics and disease-related proteomic, genomics, metabolomics and lipidomics analyses, and will not be considered in this SAP.

The analysis of all serum biomarkers for: Procollagen type I N-terminal propertide (sPINP), bone specific alkaline phosphatase (sBSAP), tartrate-resistant acid phosphatases (TRAP5b) will be described in a separate report (if analysed), and will not be considered in this SAP.

#### 2.3.2 Pharmacokinetics

The pharmacokinetics and metabolism of MIV-711 and the relationship to patient factors and concomitant medications will be described in a separate report and will not be considered in this SAP.

<sup>\*</sup>Assessments on the target knee will be used to address these other secondary objectives.

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

### 3. Study Design

This is a multicentre, randomised, placebo-controlled, double-blind, three-arm parallel, Phase IIa study to evaluate the efficacy, safety and tolerability of MIV-711 in patients with symptomatic and radiographic knee OA. A total of 240 patients with knee OA meeting the eligibility criteria and who provide written informed consent will be randomised on a 1:1:1 basis to the intervention (MIV-711 low dose 100 mg or high dose 200 mg) or placebo. Six sites distributed in 6 European countries will be used to recruit patients.

Patients who are eligible and agree to continue with the study will return for the baseline visit within 30 days of the screening visit. After baseline assessments have been completed, patients will be randomised in a 1:1:1 ratio via a central secure 24-hour randomisation service to the intervention (MIV-711) arms or the placebo-controlled arm.

- Intervention arm I: Patients will receive a once-daily 100 mg oral dose of MIV-711 for 26 weeks in addition to their current medication.
- Intervention arm II: Patients will receive a once-daily 200 mg oral dose of MIV-711 for 26 weeks in addition to their current medication.
- Control arm: Patients will receive a once-daily oral dose of matching placebo for 26 weeks in addition to their current medication.

The study consists of a screening period of approximately 4 weeks (visit 1), a baseline assessment period at visit 2, a double-blind treatment period of visit 2 through visit 8, and a follow-up period of 4 weeks (visit 9) after the last dose of study treatment is administered. Study visits for clinical assessment and questionnaires will occur at visit 2 (baseline), visit 5, visit 6, and visit 8, regardless of treatment group. The end of the study is defined as the last visit (visit 9, week 30) of the last patient or, if applicable, when the last patient has rolled over to study MIV-711-202 and having finalized visit 2 of that study.

### 3.1 Study Endpoints

The Outcome Measures in Rheumatoid Arthritis Clinical Trials (OMERACT) suggests that outcome measures for OA studies should include:

- Pain
- Function
- Quality of Life (QOL)

### 3.1.1 Primary Endpoint

The primary outcome variable is 'Pain' and will be measured using the change from

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

baseline in NRS "average" knee pain in the target knee with 7 days recall, between visit 2 (baseline) and visit 8, using a 0 to 10 NRS. The scale ranges from 0 indicating — "no pain", to 10 indicating — "pain as bad as it could be".

Other pain variables will include:

- worst target knee pain
- average contralateral knee pain
- constant and intermittent OA pain.

### 3.1.2 Secondary Endpoint

The key secondary endpoint will be the MRI of bone area in the medial femoral condyle. Bone parameters will be measured for MRIs of the target knee taken at visit 2 (baseline) and visit 8. The MRI of bone area will be assessed for the target knee.

### 3.1.3 Other Secondary Endpoints

- \*NRS e-diary assessment
- Analogsics use e-diary assessment
- \*Bone Marrow Lesions (MOAKS)
- \*Articular Cartilage (MOAKS)
- \*Osteophytes (MOAKS)
- \*Mean Cartilage thickness (Imorphics, Ltd.)
- \*Combined Bone Marrow Lesion Volume (Imorphics, Ltd.)
- Patient Reported Outcomes: to assess for pain, function, disease activity, and QOL
- Laboratory assessments for blood and urine biomarkers (Serum CTXI and urine CTXII)

### 3.1.4 Safety Endpoints

- Adverse events
- Clinical laboratory tests (hematology, clinical chemistry, and urinalysis)
- Vital signs (blood pressure, pulse, and body temperature)
- 12-lead ECGs: PR interval, QRS interval, RR interval, QT interval, and QTc interval (Bazett's correction [QTcB], Fridericia's Correction [QTcF]), heart rate
- Concomitant medication

<sup>\*</sup>These other secondary endpoints will be assessed for the target knee.

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

- Physical examination

- Rescue medication use

### 3.2 Study Population

The study population includes knee OA patients 40 to 80 years of age inclusive. The patient population fulfils the ACR criteria for OA and in addition must be radiographically confirmed as Kellgren and Lawrence (K-L) x-ray classification grade 2 or 3 and with a current average knee pain of greater or equal to 4 and less than 10 on a 1 to 10 NRS pain score. Patients must be able to provide written consent and meet all the inclusion criteria and none of the exclusion criteria.

### 3.3 Sample Size Estimation

It is planned to recruit 240 patients at 6 centers in 6 countries for this study. Recruitment will be competitive across all 6 sites.

The distribution of patients across treatment groups will be as:

MIV-711 100 mg: 80 patientsMIV-711 200 mg: 80 patients

- Placebo: 80 patients.

Details of the formal sample size calculation are provided in the protocol Section 8.7.

#### 3.4 Dose Administration

Patients will receive once-daily (OD) 100 mg or 200 mg oral dose of MIV-711, or placebo for 26 weeks in addition to their current medication. The IMP should be taken OD in the morning approximately 24 hours apart, before breakfast; breakfast can be taken approximately one hour later. The first dose is administered at the site during visit 2 (baseline). IMP should be dispensed during the visits and unused IMP returned by the patients for drug accountability at visit 5, visit 6, and visit 8. On days when the patient will visit the site the IMP must be taken at the site fasting (and not at home) and the time of the intake must be recorded in the source documents.

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

#### 3.5 Randomization

A total of 240 patients with knee OA meeting the eligibility criteria and who provide written informed consent will be randomised on a 1:1:1 basis to the intervention (MIV-711 low dose 100 mg or high dose 200 mg) or placebo.

The randomization allocation will be assigned through a centralized automated code holder that distributes the next available randomisation number on the randomisation list to the requesting site as described below.

Allocation of patients to the treatment groups will proceed through the use of an Interactive Response Technology (IRT) System [Interactive Web Response (IWR)/Interactive Voice Response (IVR) system].

The study site will obtain the randomization number and container number assignment from the IRT system. The randomization number and the date on which the randomization number was assigned will be recorded on the eCRF. Once patient screening numbers, container numbers, and randomization numbers have been assigned, they cannot be reassigned.

### 3.6 Patient Replacement

In order to perform the modified intent to treat (mITT) analysis, and to enable safety analyses, all patients who discontinue their randomised medication will be asked to still complete their follow-up visit (visit 9) as outlined in the study schedule.

Patients who withdraw from the study will not be replaced.

#### 3.7 Trial Blinding

A double-blind/masking technique will be used.

### 3.8 Protocol Deviations

The following criteria will be used to exclude a patient from the per-protocol analysis set:

- Incorrect diagnosis
- Arthroscopy in the target knee during the study period
- Missing more than 5 doses of MIV-711 (based on accountability)

Medivir Final 1.0
Protocol: MIV-711-201 22 June 2017

These criteria will be reviewed using blinded data prior to data analysis. Note: this is not an exhaustive list of deviations, these are only the deviations specified per protocol. The discussion during the BDRM will review all deviations collected at each site. All protocol deviations will be reviewed, evaluated and discussed between CRO and Sponsor before DBL.

### 3.9 Interim Analysis

No formal interim analysis that would allow early stopping of the study on the basis of demonstrating efficacy or futility is planned. Unblinded interim safety data (i.e. no efficacy analyses) will be reviewed during data monitoring committee (DMC) meetings held after 50, 100, 150 and 200 patients have completed visit 6.

#### 3.10 Extension Protocol

All patients in the current study at the participating sites included in the extension study MIV-711-202 will be given the opportunity to participate in the extension protocol provided they meet the MIV-711-202 eligibility criteria.

### 4. Study Analysis Variables

#### 4.1 Demographic and Background Variables

The following demographic and anthropometric information will be recorded at screening:

- Date of informed consent
- Medical and surgical history (including previous and current medical conditions and medications)
- Age calculated as (date of informed consent date of birth)/365.25
- Gender
- Ethnic origin
- Race
- Height (cm)
- Body weight (kg)
- Body mass index (BMI) (kg/m<sup>2</sup>)

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

### 4.2 Safety Variables

#### 4.2.1 Adverse Events

All AEs and SAEs will be recorded in the eCRF system from the date the Informed Consent Form is signed (visit 1) until the safety follow up visit (visit 9) is completed.

### 4.2.2 Clinical Laboratory Tests

Blood samples for hematology and clinical chemistry, and urinalysis assessments will be collected during all study visits: Visit 1 (screening), Visit 2 (Week 1), Visit 3 (Week 2), Visit 4 (Week 4), Visit 5 (Week 8), Visit 6 (Week 14), Visit 7 (Week 20), Visit 8 (Week 26), and Visit 9 (Week 30, follow-up).

The following safety laboratory parameters will be measured:

**Hematology:** WBC and differential, % and absolute for: neutrophils, lymphocytes, monocytes, eosinophils, basophils; hemoglobin, hematocrit, RBC, RBC indices (MCV, MCH and MCHC) and morphology, platelet count

**Chemistry:** urea nitrogen, creatinine, calcium, sodium, potassium, bicarbonate, chloride, total protein, fasting glucose, total bilirubin, direct bilirubin and indirect bilirubin, ALT, AST, alkaline phosphatase, GGT, CPK, CRP (at screening only), PTH (parathyroid hormone).

**Urinalysis**: with microscopic: specific gravity, pH, protein, glucose, ketones, nitrites, blood and leukocyte esterase

# 4.2.3 Other Laboratory Tests

- Post-menopausal determination at screening: Follicle stimulation hormone (FSH) in female patients.
- Urine Drug Screen measured at screening and Visit 5 (Week 8): Amphetamine, Benzodiazepines, THC, Cocaine, Oxycodone and Opiate.
- Serology Testing measured at screening: Hepatitis B surface antigen, total Hepatitis B core antibodies, antibodies to Hepatitis B Surface antigen, Hepatitis C virus, HIV 1 and 2.

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

# 4.2.4 Vital Signs

Vital signs (body temperature, heart rate, blood pressure, oxygen saturation) will be performed at all clinic visits prior to IMP dosing: Visit 1 (screening), Visit 2 (Week 1), Visit 3 (Week 2), Visit 4 (Week 4), Visit 5 (Week 8), Visit 6 (Week 14), Visit 7 (Week 20), Visit 8 (Week 26), and Visit 9 (Week 30, follow-up). All assessments will be collected in the supine position.

Height will be measured at visit 1 (screening) and weight will be measured at visit 1 (screening) and visit 8.

### 4.2.5 Electrocardiograms

A 12-lead ECG will be performed at all clinic visits. 12-lead serial ECGs will be recorded at visit 2 (baseline) pre-dosing and after 30 minutes, 1 hour and 2 hours post-dosing (± 10 minutes). Standard 12-lead ECG will be performed at all other visits 30 minutes after dosing (± 10 minutes).

The clinical significance of ECG results will be determined by the investigator after review of the ECG report in relation to the patient's medical history, physical examination findings, and concomitant medications.

### 4.2.6 Physical Examination

A standard complete physical examination will be performed at visit 1 (screening), visit 2 (baseline), visit 5, visit 6 and visit 8.

A targeted physical examination will be performed at visit 3, visit 4, and visit 7 assessing the following: lungs, heart, abdomen, extremity exam for the presence of peripheral oedema and lymph nodes. A standard clinical examination of both knees will be undertaken at all visits. Any clinically significant changes from visit 2 (baseline) should be recorded as AEs.

#### 4.2.7 Prior and Concomitant Medications

All concomitant medications taken during the study will be recorded with generic name, indication, daily dose, and start and stop dates of administration at each visit. For this study, prescription medicines, other than those prohibited by the study protocol are

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

permitted as concomitant medications to manage ongoing or chronic, stable medical conditions. Medications taken within 4 weeks of the screening visit will be documented as prior medication. Medication taken after the first dose of IMP will be documented as concomitant medication. Prior medications that are ongoing past Visit 2 IMP administration that involve a different dose level, frequency etc. from initial administration will be recorded as concomitant medication. Prior medications that are ongoing past Visit 2 IMP administration that do not involve a different dose level from initial administration will remain as prior medications.

The Brief Medication Questionnaire self-reported measure for the use of concomitant medication will be included at visit 5, visit 6, and visit 8.

### 4.2.8 Adherence to Study Medications

Patients will be asked to return any unused study medication at visit 5, visit 6, and visit-8 and drug accountability will be conducted.

### 4.2.9 Phone Call to Assess Safety and Tolerability

Follow-up telephone calls to assess safety and tolerability will occur 5 to 9 days after visit 2, visit 3, visit 4, visit 5, visit 6, and visit 7.

### 4.3 Pharmacodynamic Variables - Efficacy

#### 4.3.1 Pain

The primary efficacy outcome variable is 'Pain' and will be measured using the change from baseline in the average pain score for the target knee, between visit 2 (baseline) and visit 8, using a 0 to 10 NRS. The scale ranges from 0 indicating —"no pain", to 10 indicating —"pain as bad as it could be".

### 4.3.2 MRI and Imaging

The key secondary endpoint will be the change from visit 2 (baseline) to visit 8 on MRI of bone area. A secondary endpoint of interest will be the change from visit 2 (baseline) to visit 8 on MRI cartilage thickness, and the volume of bone marrow lesions. Below are the denominations of the data items that will provide the basis for bone area and cartilage thickness and bone marrow lesion volume.

- MF TAB: Area of bone in the medial femur region, MF
- CM\_FEMUR\_THCTAB: Average thickness of cartilage in the central medial femur region

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

- CM\_TIBIA\_THCTAB: Average thickness of cartilage in the central medial tibia region
- TOTAL\_BML\_VOLUME: Combined volume of all BML regions

Other secondary endpoints will include the analysis of MRIs using MOAKS scoring.

MRI assessment using MOAKS scoring will be used to assess the following features, as provided by PAREXEL MRI:

- Bone Marrow Lesions (BMLs) and cysts. This involves 15 subregions graded for BML size (including ill-defined lesion and cysts) measuring the total volume of the subregion occupied by BML(s). Grade 0= none, grade 1 < 33% of subregional volume, grade 2 = 33 to 66% of subregional volume and grade 3 > 66% of subregional volume.
- Articular Cartilage: This involves 14 articular cartilage regions graded for size of any cartilage loss (including partial and full thickness loss) as a percentage of surface area as related to the size of each individual region surface and percentage of loss in this subregion that is full-thickness loss.
- Osteophytes: This involves 12 sites scored for presence and size of osteophytes. Grade 0=none, Grade 1= small, Grade 2 = medium, Grade 3 = large.

The specific subregrions associated with the above three groups of MOAKS scoring are outlined in the table below:

| Bone Marrow Lesions (BMLs) and cysts | Articular Cartilage | Osteophytes |
|---|---|---|
| Medial Patella | Medial Patella | Superior Patella |
| Lateral Patella | Lateral Patella | Inferior Patella |
| Medial Femur Trochlea | Medial Femur Trochlea | Medial Patella |
| Medial Femur Central | Medial Femur Central | Lateral Patella |
| Medial Femur Posterior | Medial Femur Posterior | Medial Femur Trochlea |
| Lateral Femur Trochlea | Lateral Femur Trochlea | Medial Femur Central |
| Lateral Femur Central | Lateral Femur Central | Medial Femur Posterior |
| Lateral Femur Posterior | Lateral Femur Posterior | Lateral Femur Trochlea |
| Medial Tibia Anterior | Medial Tibia Anterior | Lateral Femur Central |
| Medial Tibia Central | Medial Tibia Central | Lateral Femur Posterior |
| Medial Tibia Posterior | Medial Tibia Posterior | Tibia Medial |
| Subspinous | Lateral Tibia Anterior | Tibia Lateral |
| Lateral Tibia Anterior | Lateral Tibia Central | |
| Lateral Tibia Central | Lateral Tibia Posterior | |
| Lateral Tibia Posterior | | |

Bone Marrow Lesions (BMLs) and cysts: The 15 subregions will be assessed for:

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

- Size of BML
- Number of BMLs
- Percentage that is BML

Articular Cartilage: The 14 subregions will be assessed for:

- Size of any cartilage loss
- Percentage of Full Thickness Loss

### 4.3.3 Patient Reported Outcomes (PRO)

Patient-reported outcomes will be recorded using questionnaires at visit 2 (baseline) and at visit 5, visit 6, and visit 8. These PRO data will be used as measures of pain, function and disease activity.

### 4.3.3.1 NRS Scores - Knee Pain and Function in the Last Week

For the purposes of the questions below, the <u>target knee</u> is defined as the knee studied in this trial. Pain in your knee relates to any knee symptom you may experience for example pain or aching.

The scale ranges for NRS pain scores range from 0 indicating —"no pain", to 10 indicating —"pain as bad as it could be". The NRS scales will be used to assess for:

- 1) NRS question 1: NRSPTO (Primary Endpoint). On average, how would you rate the overall pain severity in your <u>target</u> knee over the last week (7 days)?
- 2) NRS question 2: NRSPAINW. How would you rate your <u>worst</u> pain severity in your target knee over the last week (7 days)?
- 3) NRS question 3: NRSPAINS. On average, how would you rate the overall pain severity in your <u>other</u> knee over the last week (7 days)?
- 4) NRS question 4: NRSACT. Over the last week (7 days), how active do you think your target knee arthritis has been?
- 5) NRS question 5: NRSSAT. Over the last week (7 days), how satisfied have you been with your target knee function?

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

For purposes of this SAP NRS question 4 refers to the patients "Global Assessment Score".

#### 4.3.3.2 ICOAP Scores

Intermittent and constant osteoarthritis pain (ICOAP): an 11-item tool designed to assess constant and intermittent pain. Higher scores indicate worse constant and intermittent pain. The items assessed include:

- IP1- How intense has constant knee pain been
- IP2-Constant knee pain affecting sleep
- IP3-Constant knee pain quality of life
- IP4-Frustrated by your constant knee pain
- IP5-Upset by your constant knee pain
- IP6-Intensity of pain that comes and goes
- IP7-Frequency pain that comes and goes
- IP8-Pain comes and goes affecting sleep
- IP9-Pain comes and goes quality of life
- IP10-Frustration pain that comes and goes
- IP11-Upset pain that comes and goes

#### 4.3.3.3 WOMAC Scores

Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) 3.1: a 24-item OA - specific, tri-dimensional self-administered questionnaire, for assessing health status and health outcomes in OA of the knee. Using an 11-box NRS scale, higher scores indicate worse pain, stiffness and physical function. Items assessed include:

- WOMAC1-Pain walking on a flat surface
- WOMAC2-Pain going up or down stairs
- WOMAC3-Pain at night while in bed
- WOMAC4-Pain sitting or lying down
- WOMAC5-Pain while standing
- WOMAC6-Stiffness after first woke up in morning
- WOMAC7-Stiffness sitting or lying down
- WOMAC8-Difficulty When going down the stairs
- WOMAC9-Difficulty When going up the stairs
- WOMAC10-Difficulty Getting up from a sitting
- WOMAC11-Difficulty While standing

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

- WOMAC12-Difficulty When bending to the floor
- WOMAC13-Difficulty Walking on a flat surface
- WOMAC14-Difficulty Getting in or out of a car
- WOMAC15-Difficulty While going shopping
- WOMAC16-Difficulty When putting on your socks
- WOMAC17-Difficulty When getting out of bed
- WOMAC18-Difficulty When taking off your socks
- WOMAC19-Difficulty While lying in bed
- WOMAC20-Difficulty Getting in or out of bath
- WOMAC21-Difficulty While sitting
- WOMAC22-Difficulty Getting on or off toilet
- WOMAC23-Difficulty Performing heavy duties
- WOMAC24-Difficulty Performing light duties

#### 4.3.3.4 OMERACT Scores

Osteoarthritis Research Society International (OARSI)-OMERACT Responder index [2, 3] will be calculated using the WOMAC pain and function subscales and the patient's global assessment score. A responder will be defined as any subject that satisfies one of the following two overall conditions:

CASE 1. Improvement in pain or function  $\geq$ 50% and absolute change  $\geq$ 20

CASE 2. Improvement in at least two of the following conditions:

- 1. pain >20% and absolute change >10
- 2. function  $\geq 20\%$  and absolute change  $\geq 10$
- 3. patients' global assessment  $\geq 20\%$  and absolute change  $\geq 10$

Higher scores indicate worse pain, stiffness and physical function so that an "improvement" is only concerned with negative changes (or decreases) from baseline. Positive increases in scores relative to baseline suggest a worsening of pain (scores increasing over time suggests pain is increasing in severity over time).

### 4.3.3.5 Global Improvement Scores

Global improvements in knee problem, knee pain and knee function (Ability to use knee) recorded on a 6-point likert scale at visit 5, visit 6, and visit 8 only: (completely better, much better, better, no change, worse, much worse)

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

### 4.3.3.6 Quality of Life

At visit 2 (baseline) and visit 8: EuroQol -5 Dimensions (EQ-5D-5L) - a generic measure of self-reported health status. Items assessed include:

- Usual Activities
- Anxiety/Depression
- Self-Care
- Pain/Discomfort
- Mobility
- Health Rating

### 4.3.3.7 Brief Medication Questionnaire

The Brief Medication Questionnaire is a self-reported measure for the use of concomitant medication and will be administered at visit 5, visit 6, and visit 8. Items assessed include:

- How much did you take each time
- How many days did you take it
- The dosage times are inconvenient
- How many times per day did you take it
- It is hard to get my refill on time
- How many times did you miss taking it
- It is hard to open the container
- Hard to read the print on the container
- For what reason were you taking it
- It is hard to remember all doses
- Stop taking meds since(V5) or (V6, V8)
- Medication Name

### 4.3.3.8 E-Diary Assessment of NRS and Analgesic Use

In an e-diary format, a patient knee pain diary (NRS) and analgesia questionnaire will be completed daily every 12 hours (AM, PM) during three two-week periods prior to visit 2 (baseline), visit 6 and visit 8. Baseline will be defined as the last observation prior to the first dose of investigational product. The assessments in the e-diary comprise:

- Average overall knee pain severity in the target knee over the past 12 h (0 -10 NRS)
- Adherence to usual analgesics regimen:
  - o Has patient taken any pain medication over last 12 hours? (Yes, No).

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

- Classify your pain medication usage over the last 12 hours: (More than normal, Normal, Less than normal)
- Intake of IMP (note: the e-diary device is kept by the patients for the full duration of the study, intake of IMP will be registered daily throughout the study)

### 4.3.4 Secondary Efficacy Parameters

#### 4.3.4.1 Biomarkers

Secondary Endpoints: Blood and urine samples for the analysis of secondary and exploratory bone and cartilage markers of relevance for OA disease for analysis of serum CTX-I and urinary CTX-II biomarkers will be taken at visit 2 (baseline) and visit 4, visit 6, visit 8, and visit 9.

- urinary CTX-II biomarkers
- serum CTX-I

### 4.3.4.2 Other Imaging Assessments

K-L scoring based on target knee radiographs no older than 12 months is required to assess inclusion criterion 3.

At visit 2 (baseline) and visit 8, MRI acquisition will be performed on the target knee for measurement of bone area, cartilage thickness and BML volume.

### 4.4 Analysis Populations

### 4.4.1 Intent-to-Treat Population (ITT)

All randomised patients in the treatment group to which they were randomised, regardless of whether treatment was received as planned.

### **4.4.2 Modified Intent-to-Treat Population (mITT)**

mITT is the full analysis set (FAS) consisting of all patients having both a baseline and at least one post-baseline value for the primary variable (NRS pain score).

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

### 4.4.3 Per Protocol Population (PPS)

Those patients who adhered to the treatment regimen of the program to which they were allocated, provided sufficient assessment of primary outcomes, and did not violate the study protocol in any substantial way.

### 4.4.4 Safety Analysis Population (SAF)

The safety analysis population will include all patients receiving at least one dose of either MIV-711 or placebo. These patients will be analyzed according to treatment actually received.

#### 5. General Considerations for Data Presentations

In this study IMP refers to any amount of the treatments defined in section 3.4, regardless of the time or period of administration.

Data for all enrolled patients who receive at least one dose of IMP will be presented in the data listings.

A patient who is enrolled but does not receive IMP will be included in those data listings for which they have data but will be excluded from all data summaries. Data summaries will only include those patients that receive IMP.

For those listings or data summaries where baseline and change from baseline measurements will be presented, unless stated otherwise, the baseline assessment to be used for calculating change from baseline will be the last valid assessment prior to first dose administration.

All pre- and post-dose assessments including unscheduled assessments will be included in the data listings. For unscheduled assessments collected pre-dose, the last assessment taken for a time point will be used in the data summaries (summary tables, figures, and statistical analysis); for all post-dose time points, the original assessment for any given time point will be used in the data summaries (summary tables, figures, and statistical analysis).

For summaries of safety data continuous variables will be summarized using descriptive statistics including: number of observations (n), mean (arithmetic), median, standard deviation (SD), minimum, and maximum. Frequencies and percentages will be used for summarizing discrete (categorical) data. In summaries for safety the denominator for all percentages will be the number of patients in a given treatment group.

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

Safety and efficacy data that are reported as missing will be excluded from all descriptive and non-descriptive data analysis. There will be no imputation of any data. Observations that might be considered spurious (extreme relative to the majority of the data) will not be altered or removed from any presentation of the data, including the calculation of summary statistics (means, medians, etc.), unless approved by the sponsor.

For data listings, all raw data will be reported/displayed exactly as provided. For summaries of quantitative safety data, the minimum and maximum value will be reported exactly as the raw data are reported; measures of central tendency (means, medians) will be reported to one more decimal place than the raw data; measures of variance (SD) will be reported to two more decimal places than the raw data.

Unless stated otherwise there will be no adjustment for multiple comparisons. All statistical tests will be one-sided and will be performed at the 5% level of significance (Type I error =0.05).

In all data persentations 'Treatment' will be defined as consisting of the three protocol defined categories: 200 mg, 100 mg, placebo. Listings will include all patients and will be sorted by treatment, patient number, and time point (where applicable). In all listings treatment will be grouped in the order: 200 mg, 100 mg, placebo. All derived data used in a data summary or statistical analysis will be listed.

#### 5.1 Software

All statistical analyses will be performed using Statistical Analysis Software (SAS®) (SAS® Institute Inc., Cary, North Carolina, United States of America [USA]) Version 9.2 or higher.

#### 6. Patient and Treatment Information

#### 6.1 Patient Disposition

The completion status, date of completion or discontinuation, the reason for discontinuation, and the study day of withdrawal will be listed. The number of patients enrolled and the frequency and percentage of patients completing the study, patients withdrawing early, and primary reason for withdrawal will be summarized by treatment and overall. Also included in this summary will be the numbers of patients in each of the analysis populations: ITT, mITT, PPS.

Per protocol patients will take IMP until V8 and then they have a safety follow up visit (V9) 4 weeks after last IMP dose. If a patient is withdrawn IMP is stopped but the patient

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

is still asked to come for the safety follow up visit (V9) 4 weeks after last IMP. Some patients are withdrawn but refuse or are unable to attend the safety follow up visit (V9) 4 weeks later.

### 6.2 Patients Excluded from Analysis Populations

Each patient excluded from one of the analysis populations will be listed along with the reason for their exclusion.

### 6.3 Eligibility Criteria

All enrolled patients who did not meet an inclusion criterion and all enrolled patients who met an exclusion criterion will be listed.

#### **6.4** Exclusion Tests

Results of the exclusion tests will be listed. These will include laboratory tests performed prior to dosing for: FSH testing, serology, and urine drug screen.

#### 6.5 Protocol Deviations

Deviations from the protocol including violations of inclusion/exclusion criteria will be assessed as minor or major in cooperation with the sponsor. Major deviations from the protocol may lead to the exclusion of a patient from the Per Protocol Set (PPS). Deviations will be defined prior to unblinding. All reported protocol deviations will be listed.

#### 6.6 Demographic Data

Demographic and baseline characteristics will be evaluated for the ITT and for the PPS. Demographic information will be listed. Descriptive statistics will be obtained for the continuous variables: height, age, BMI, and body weight and presented overall. Frequencies and percentage of patients will be tabulated for the categorical variables ethnicity, race, and gender.

### 6.7 Medical History

Medical and surgical history data recorded prior to dosing will be listed for each patient. Medical history will be coded using the MedDRA (Version 18.1).

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

Only those body systems where a condition or abnormality has been reported will be listed.

#### 6.8 Prior and Concomitant Medication

Prior and concomitant medications will be coded using WHO Drug (September 2015 version). These medications will be classified by Anatomical Therapeutic Chemical (ATC) categories.

Prior and Concomitant Medications will be listed by patient.

Summary tables of the number of percentage of patients by treatment and ATC classification will be provided for prior and concomitant medications.

#### 6.9 Dose Administration

Information collected per the dose administration CRF will be listed including patient number, treatment, visit, and the date and time of administration as well as the dose form, route of administration, number of capsules dispensed and number of capsules returned.

The number and percentage of patients who received IMP will be summarized for each on site visit and by treatment. Descriptive statistics will be used to summarize drug accountability as the number of capsules returned for each on site study visit by treatment.

Compliance will be derived as the number of days patient was exposed to IMP. 100% compliance will be considered for dosing during the period Visit 2 to Visit 8. The number of capsules used will be derived as the number of capsules dispensed minus the number of capsules returned. Subjects with less than 100% compliance will be identified among those who have results for "Reason not all unused Capsules returned".

# 7. Pharmacodynamic Analysis - Efficacy

The primary and secondary efficacy analysis will be based on the mITT population.

#### 7.1 NRS Pain Data

NRS data for knee pain will be listed for each patient, treatment, and time point. NRS results will be shown for the following:

• Primary endpoint: Amount of pain severity in the target knee last week (SDTM: Overall pain severity in target knee

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

- Global Assessment Score: How active has the target knee arthritis has been in the past week (SDTM: How active was target knee arthritis)
- Satisfaction with target knee function (SDTM:How satisfied are you with target knee function)
- Worst pain severity in target knee (SDTM: Worst pain severity in target knee)
- Overall pain severity in other knee (SDTM: Overall pain severity in other knee)

Change from baseline will be derived for each of the above NRS pain scores. These changes from baseline scores will be descriptively summarized by visit and treatment. Frequency tables by treatment will be used to summarize the number and percent of patients in each of the categories observed for:

- Duration of Knee Pain Past 12 Months: Within the last 7 Days, Days 8-30, Days 31-92, More than 92 Days
- Onset of Knee Pain: Within the last 12 months, 1 to 5 years, 5 to 10 years, More Than 10 years

Results for duration and onset of knee pain will be listed for each patient.

Graphical presentation of the observed and change from baseline NRS pain scores will include:

- Mean ± 95% CI Profiles of Observed NRS Scores by Treatment, mITT Population
- Mean ± 95% CI Profiles of Change From Baseline NRS Scores by Treatment, mITT Population

### 7.2 Statistical Analysis of the NRS Pain Data

To assess the sensitivity of the statistical analysis to the choice of analysis set, the primary efficacy analysis described below will be considered for both the mITT and the PPS populations.

The primary hypothesis of this study is that MIV-711 will reduce pain in patients with moderate knee osteoarthritis diagnosed based on symptomatic and radiologic criteria. To statistically test this hypothesis, a linear mixed model via SAS PROC MIXED based on the FAS (mITT). The model will include fixed factors for treatment, time (measured in weeks), the interaction for treatment-by-time, baseline analgesic user (Yes/No), and random effect for clinical site. The baseline NRS score will be included as a covariate for adjustment.

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

Patients considered pain medication users at baseline will be identified via concomitant medication analysesic usage. Pain medication users will include any patient exposed to a prescribed analysesic at time of first IMP intake and the medication was ongoing at the time of visit 2.

The dependent variable in the linear model is the change from baseline NRS pain score. Separate mixed model analyses will be considered for each of the change from baseline NRS pain scores.

- Primary endpoint: Amount of pain severity in the target knee last week (SDTM: Overall pain severity in target knee
- Global Assessment Score: How active has the target knee arthritis has been in the past week (SDTM: How active was target knee arthritis)
- Satisfaction with target knee function (SDTM:How satisfied are you with target knee function)
- Worst pain severity in target knee (SDTM: Worst pain severity in target knee)
- Overall pain severity in other knee (SDTM: Overall pain severity in other knee)

In this analysis the contrast of primary interest is the treatment difference (active versus placebo) at visit 8 week 26. LSmeans at visit 8 for the change from baseline score will be reported from the mixed model. LSmeans for the overall effect of treatment, estimates of the pair-wise treatment differences, two-sided 95% confidence intervals (CI), and p-value (one-sided) will be provided.

The following SAS code maybe used as reference:

```
PROC MIXED data=;
CLASS patient treatment week;
MODEL NRS_chg= NRS_baseline treatment week treatment*week baseline_conmed_pain_use/
DDFM=KR;
RANDOM site;
REPEATED week / SUBJECT=patient TYPE=UN;
LSMEAN treatment*week treatment / diff CL ALPHA=0.1;
RUN;
```

In an alternate sensitivity analysis of the primary endpoint (Amount of pain severity in the target knee last week) that could be considered as applicable, the linear model described in this section would include the PRO for e-diary analgesic use (Yes, No) as an additional independent factor. This analysis would be considered only if baseline pain medication usage could not be adequately identified via the concomitant medication records. The effect of whether or not a patient was an analgesic user at baseline as defined by the e-diary would then be considered as the additional factor.

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

### 7.2.1 Multiplicity Adjustment for the Primary Endpoint

For the primary endpoint, change from visit 2 (baseline) to visit 8 in NRS pain score, the Type I error for the tests of the two doses will be protected by performing a fixed-sequence multiple-testing procedure. The order of steps is defined below:

Step 1. 200 mg versus placebo

Step 2. 100 mg versus placebo

To adjust for the multiple testing of two doses, the second step will only be considered as confirmatory providing the previous step is significant at a one-sided 5%-level (p<0.05). If the previous step is not significant, the analysis of the following step will be considered descriptive.

### 7.2.2 Visualizations for the Primary Endpoint

Mean profiles for treatments (MIV-711) will be compared with placebo for each treatment as well as the difference from placebo treatment, as obtained from the change from baseline NRS score estimated least squares means. The difference from placebo in least squares means obtained from the above mixed model (section 7.2) will be presented in the following figures:

- NRS Change From Baseline (LSMean Difference ± 95% CI) Difference from Placebo by Treatment and Time Point, mITT Population
- NRS Change From Baseline (LSMean Difference ± 95% CI) Difference from Placebo by Treatment and Time Point, PPS Population

### 7.3 Key Secondary Analysis: MRI of Bone Area in Target Knee

The observed and change from baseline of the MRI of the bone area of the medial femur for the target knee will be listed for each patient and descriptively summarized by treatment and visit.

#### 7.3.1 Statistical Analysis of the MRI of Bone Area in Target Knee

As the key secondary analysis of efficacy, the change from baseline in the MRI of bone area in the target knee will be analysed using the same statistical model described in

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

Section 7.2 above. This analysis will be based on the mITT population. Results will be summarized.

Mean profiles for treatments (MIV-711) will be compared with placebo by plotting the difference from placebo using the change from baseline MRI bone area score:

MRI of Bone Area Change From Baseline (LSMean Difference ± 95% CI)
 Difference from Placebo by Treatment and Time Point, mITT Population

### 7.4 Secondary Analysis: MRI of Cartilage Thickness in Target Knee

The observed and change from baseline of the MRI of the cartilage thickness for the target knee will be listed for each patient and descriptively summarized by treatment and visit. Source data for these analyses will be obtained from:

- CM\_FEMUR\_THCTAB: Average thickness of cartilage in the central medial femur region
- CM\_TIBIA\_THCTAB: Average thickness of cartilage in the central medial tibia region

### 7.4.1 Statistical Analysis of the MRI of Cartilage Thickness in Target Knee

As a secondary analysis of efficacy, the change from baseline in the MRI of cartilage thickness in the target knee will be analysed using the same statistical model described in Section 7.2 above. This analysis will be based on the mITT population. Results will be summarized.

Mean profiles for treatments (MIV-711) will be compared with placebo by plotting the difference from placebo using the change from baseline MRI cartilage thickness score:

MRI of Cartilage Thickness Change From Baseline (LSMean Difference ± 95% CI) Difference from Placebo by Treatment and Time Point, mITT Population

#### 7.5 Secondary Analysis: MRI of total BML Volume in Target Knee

The observed and change from baseline of the MRI of the total bone marrow lesion volume for the target knee will be listed for each patient and descriptively summarized by treatment and visit. Source data for these analyses will be obtained from:

- Total BML Volume

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

# 7.5.1 Statistical Analysis of the MRI of Total BML Volume in Target Knee

As a secondary analysis of efficacy, the change from baseline in the MRI of total bone marrow lesion volume in the target knee will be analysed using the same statistical model described in Section 7.2 above. This analysis will be based on the mITT population. Results will be summarized.

Mean profiles for treatments (MIV-711) will be compared with placebo by plotting the difference from placebo using the change from baseline MRI cartilage thickness score:

MRI of Total BML Volume Change From Baseline (LSMean Difference ± 95% CI) Difference from Placebo by Treatment and Time Point, mITT Population

### 7.6 Analysis of Other Secondary Imaging Assessments

Other secondary imaging variables will be listed for each patient and descriptively summarized by treatment and visit. These other secondary imaging variables will include:

#### **MOAKS** Variables

- Bone Marrow Lesions (BMLs) and cysts
  - o Size of BML: 0='None', 1='<33%', 2='33-66%', 3='>66%',9='Not Evaluable'
  - o Number of BMLs: scored 9 to 99
  - Percentage that is BML: 0='None', 1='<33%', 2='33-66%', 3='>66%', 9='Not Evaluable'
- Articular Cartilage
  - Size of any Cartilage Loss: 0='Normal', 1='<10% Area', 2='10-75% Area', 3='>75% Area', 9='Not Evaluable'
  - o Percentage Full Thickness Loss: 0='Normal', 1='<10% Region', 2='10-75% Region', 3='>75% Region', 9='Not Evaluable'
- Osteophytes: 0='None', 1='Small', 2='Medium', 3='Large', 9='Not Evaluable'

For the MOAKS imaging variables collected quantitatively the change from baseline score will be derived and descriptively summarized by treatment and visit. For MOAKS variables with categorical response, the number and percentage of subjects in each treatment for each category will be summarized.

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

# 7.7 Analysis of Other Patient Reported Outcomes (PROs)

### 7.7.1 Intermittent and Constant Osteoarthritis Pain (ICOAP) Knee Version

The observed raw ICOAP scores will be listed by treatment and visit for each patient.

The observed results for the intermittent and constant osteoarthritis pain (ICOAP) score will be transformed to a 0-100 scale for analysis. The following methods will be used to transform the ICOAP scores:

### Constant pain subscale

To calculate the Total constant pain subscale, sum the scores within each time point for items IP1 through IP5. Maximum constant pain score ranges from 0 to 20.

This score can be transformed to a score out of 100 using the following formula:

(Total constant pain score / 20) x 100

### *Intermittent pain subscale*

To calculate the total intermittent pain subscale, sum the scores within each time point for items IP6 through IP11. Maximum intermittent pain subscale ranges from 0 to 24. This score can be transformed to a score out of 100 using the following formula:

(Total intermittent pain score / 24) x 100

### Total pain score

To calculate the total ICOAP score, sum the constant and intermittent pain subscales within each time point. Maximum total pain score ranges from 0 to 44. This score can be transformed to a score out of 100 using the following formula:

(Total pain score / 44) x 100

The three transformed ICOAP scores (Constant Pain, Intermittent Pain, and Total Pain) will be listed by patient for each scheduled time point. Change from baseline will be derived for each of these transformed ICOAP scores. The observed and change from baseline values for these three transformed ICOAP scores will be listed and the change from baseline values will be descriptively summarized by treatment and time point. Figures of the mean change from baseline ICOAP response, using each transformed ICOAP score, will be used to visualize the behavior of the ICOAP response over time:

• ICOAP Change From Baseline by Treatment and Time Point, mITT Population

 Medivir
 Final 1.0

 Protocol: MIV-711-201
 22 June 2017

### 7.7.2 Analysis of the WOMAC

The observed WOMAC scores for pain, stiffness, and physical function will be listed. Change from baseline scores will be derived for each WOMAC item, listed by patient and descriptively summarized by treatment and visit.

Mean profiles for treatments (MIV-711) will be compared with placebo by plotting the change from baseline WOMAC score:

- WOMAC Pain Score Mean Change From Baseline (95% CI) by Treatment and Time Point, mITT Population.
- WOMAC Stiffness Score Mean Change From Baseline (95% CI) by Treatment and Time Point, mITT Population
- WOMAC Difficulty Score Mean Change From Baseline (95% CI) by Treatment and Time Point, mITT Population

### 7.7.3 (OARSI)-OMERACT Responder Criteria

The following steps will be used to derive OARSI-OMERACT response (Yes, No). This analysis will use the PROs from the WOMAC pain data, the WOMAC Function data, and the patient global assessment NRS observed at Visit 2 and Visit 8. It is expected Visit 8 will be the last 'on-treatment' visit for each subject.

#### Step 1. Derive Total Scores:

- a) Total WOMAC Pain (Sum of 5 questions): For each subject and each scheduled time point derive a total score by summing over all 5 pain responses. For each subject this will provide a total WOMAC Pain score out of 50 for each protocol scheduled time point. Denote this new variable in the data set as 'WOMAC Pain 50'.
- b) Total WOMAC Function (Sum of 17 questions): For each subject and each scheduled time point derive a total score by summing over all 17 difficulty responses. For each subject this will provide a Total WOMAC Function score out 170 for each protocol scheduled time point. Denote this new variable in the data set as 'WOMAC Func 170'.
- c) Patient Global Assessment (NRS question 4: Over the past week, how active do you think your knee arthritis has been?). Use this score as is, scored out of 10.

Step 2. Transform the three scores from Step 1 to create three new scores, each out of 100:

a) Transformed WOMAC Pain Score: WOMAC PAIN 100 = WOMAC Pain 50 ⊠ 2.

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

- b) Transformed WOMAC Function Score: WOMAC FUNC 100 = WOMAC Func 170 ÷1.7.
- c) Transformed Global Assessment Score:
  NRSACT\_100 = (Global Assessment Score ) ⊠ 10.

Step 3. Comparing Visit 8 against Visit 2: Use the transformed scores from step 2 to derive change between baseline and percentage change from baseline scores.

Denote the change from baseline scores as:

- CHG WOMAC PAIN 100
- CHG WOMAC FUNC 100
- CHG NRSACT 100

Denote the percentage change from baseline scores as:

- PCHG WOMAC PAIN 100
- PCHG WOMAC FUNC 100
- PCHG\_NRSACT\_100

Percentage change from baseline will be calculated as: ((Visit 8 Score – Visit 2 Score) ÷ Visit 2 Score) ⊠ 100

The total scores and the transformed scores for each of WOMAC pain, WOMAC physical function, and global assessment will be listed by patient and visit along with their change from baseline scores and percentage change from baseline scores. Change from baseline scores will be presented for Visit 8 only. Percentage change from baseline scores will be derived from visit 2 and visit 8 data only.

Step 4. Derive Responder OARSI-OMERACT (Yes, No): In all derived scores, low values are associated with less severe pain (0 = no pain) and high scores are associated with more severe pain (100 = worst pain). In assessing for a positive OMERACT response, patient improvement (Response = Yes) is associated with decreases (negative changes) from baseline and (negative) percentage (changes) decreases from baseline. The different criteria are quantified in the tables below.

Case 1: using the change from baseline and percentage change from baseline scores for WOMAC pain and WOMAC function (from step 3), an OMERACT responder will be flagged as 'Yes' if either of the following 2 criteria are satisfied:

| | | Percentage | |
|----------|---------------|---------------|-----------|
| | Decrease from | Decrease from | OMERACT |
| Criteria | Baseline | Baseline | Responder |
Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

| 1 | WOMAC Pain | ≥ 20 | and | ≥ 50% | Yes |
|---|----------------|------|-----|-------|-----|
| 2 | WOMAC Function | ≥ 20 | and | ≥ 50% | Yes |

Case 2: using the change from baseline and percentage change from baseline scores for WOMAC pain, WOMAC function, and global assessment score (from step 3), an OMERACT responder will be flagged as 'Yes' if <u>at least</u> 2 of the following 3 criteria are satisfied:

| Criteria | | Decrease<br>from<br>Baseline | | Percentage<br>Decrease from<br>Baseline | OMERACT<br>Responder |
|---|---|---|---|---|---|
| 3 | WOMAC Pain | ≥ 10 | and | ≥ 20% | Yes |
| 4 | WOMAC Function | ≥ 10 | and | ≥ 20% | Yes |
| 5 | Global Assessment NRS | ≥ 10 | and | ≥ 20% | Yes |

A subject is a 'Yes' responder if either of criteria 1 or 2 are satisfied. If neither criteria 1 or 2 are satisfied, criteria 3, 4 and 5 will be checked.

A listing will be created that presents each patient's responder status by treatment. Included in this listing will be the associated change from baseline and percent change from baseline values.

The number and percentage of subjects with responder status will be summarized by treatment.

#### 7.7.4 Global Improvements

Global improvements in knee problem, knee pain and knee function that were recorded on a 6-point likert scale: completely better, much better, better, no change, worse, much worse.

Descriptive tables will be used to summarize the number and percentage of each global improvement response for each treatment group by time point. All data will be listed for each patient.

### 7.7.5 Quality of Life PRO – EQ-5D-5L

Observed results from the EQ-5D-5L will be listed for each patient.

This will include results from the 5 dimensions: mobility; self-care; usual activity; pain or discomfort; and anxiety or depression, in addition to the reported health rating score.

Change from baseline scores will be derived for each QOL response as Visit 8 Week 26

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

versus Visit 2 Day 1. The change from baseline scores will be summarized using descriptive statistics by treatment group. The observed mean scores with 95% CI will be plotted by treatment and time point to visualize the QOL response over time.

### 7.7.6 E-diary for Patient Pain

All data collected in e-diary format, will be listed for each patient.

Data permitting summary tables by treatment and time point will be provided for the e-diary information reported for NRS scores and pain medication usage.

Separate summary tables will be provided for AM and PM response as well as a table for overall 24 hour response. The overall summary will use the mean of the AM and PM NRS scores provided for each visit, to obtain one record for that visit.

The number and percentage of patients with 'Yes/No' response to pain medication usage on the e-diary will be provided separately for AM, PM as well as for 24 hours overall. For the overall table, at least one 'Yes' response, either for the AM or the PM response, will be interpreted as a 'Yes' response over the 24 hours.

The number and percentage of patients with each pain medication usage response ('More than Normal', 'Normal', 'Less than normal') will be summarized by treatment and visit, with separate summaries for AM and PM response.

Data permitting the average NRS e-diary score will be visualized using a plot of mean NRS response by treatment and time point. Separate figures will be provided for the AM and PM NRS scores as well as overall 24 hours for each visit. For the overall figure the mean of the AM and PM NRS scores will be used to obtain 1 record at each visit prior to computing descriptive statistics.

### 7.7.7 Biomarkers from Serum and Urine Samples

The serum CTX-I and urinary CTX-II biomarkers will be presented in data lisitings by subject and time point and in descriptive summary tables by treatment and time point. Figures of mean response over time with +/- 95% CI will be used to visualize their distribution over time for each treatment.

Time-Integrated-Concentrations (TIC) will be derived for each serum CTX-I and urinary CTX-II biomarkers. For each biomarker the mean TIC value and the standard deviation (SD) of the TIC will be derived. For each biomarker a Z- score will be derived by subtracting the mean and dividing by SD. TIC results and associated Z-scores will be listed for each subject.

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

#### 8. Safety Analysis

All safety analyses will be based upon the SAF. If one or more patients received incorrect IMP, these data will also be presented for the SAF.

#### 8.1 Adverse Events

All AEs reported will be coded and classified according to MedDRA version 18.1.

A treatment-emergent AE (TEAE) will be defined as an AE that begins or that worsens in severity after IMP has been administered.

Non-treatment emergent adverse events (NTEAE): AEs that occurred before the administration of IMP and did not worsen in severity or relationship after exposure to IMP.

All AE data as captured on the CRF will be listed by patient. All serious AEs (SAEs) will be listed. A listing of all AEs leading to treatment discontinuation will be presented.

Unless specified otherwise, all adverse event summaries will include the TEAEs only and adverse event summary counts of AEs will be the number of patients reporting adverse events and not the number of events reported. The number and percentage of patients with adverse events will be tabulated by body system and preferred term for each treatment. A patient with multiple adverse events within a body system is only counted once towards the total of that body system. If the same AE (preferred term) is reported several times for the same patient, it will only appear once for that specified treatment in the summary tables.

For patients with multiple adverse events of the same preferred term and of different severities, the AE with the highest assessment of severity will be used in the summaries presented by severity.

Presentations of AEs (tables and listings) will be by treatment defined by the dose level of MIV-711 and placebo.

A general summary of all treatment-emergent adverse events will show the number and percentage of patients, as well as the number of events, according to the following categories:

- All treatment emergent adverse events
- 'Related' treatment emergent adverse events
- Mild treatment emergent adverse events
- Moderate treatment emergent adverse events
- Severe treatment emergent adverse events

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

- Serious treatment emergent adverse events
- Treatment emergent adverse events leading to early termination
- Deaths

Other summary tables for adverse events will include:

- Number and Percentage of Patients with Treatment Emergent Adverse Events by System Organ Class, Preferred Term, and Treatment
- Number and Percentage of Patients with Treatment Emergent Adverse Events 'Related to IMP' by System Organ Class, Preferred Term, Severity, and Treatment.
- Number and Percentage of Patients with Treatment Emergent Adverse Events 'Not Related to IMP' by System Organ Class, Preferred Term, Severity, and Treatment.
- Number and Percentage of Patients with Serious Treatment Emergent Adverse Events by System Organ Class, Preferred Term, and Treatment
- Number and Percentage of Patients with Treatment Emergent Adverse Events Leading to Discontinuation by System Organ Class, Preferred Term, and Treatment

### 8.2 Clinical Safety Laboratory Tests (Hematology, Chemistry, Urinalysis)

### **8.2.1** Hematology and Chemistry

A by-patient listing of all observed chemistry and hematology laboratory data will be provided. Laboratory results outside the normal range will be flagged. The abnormal values will be flagged with 'L' (low) for values below the lower limit of the laboratory's normal range or 'H' (high) for values above the upper limit of the laboratory's normal range. Abnormal values will be graded as not clinically significant (NCS) or clinically significant (CS). Clinically significant laboratory results will be included in the AE listings.

The observed values of all safety laboratory assessments for clinical chemistry and hematology will be summarized using descriptive statistics showing the number of observations (n), mean, median, SD, minimum, and maximum value. Table summaries will be presented by treatment and time point.

Baseline values for all clinical chemistry and hematology parameters will be categorized as being below the normal range (Low), within the normal range (Normal), and above the normal range (High). Shift from baseline tables will present the frequency and percentage of patients who have observations that are Normal, Low, or High. Shift tables will be presented by treatment group for values shifting from Day -1 to the maximum and the minimum post-dose value.

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

All hematology, chemistry, and coagulation, laboratory parameters noted in Section 4.2.2 of this SAP will be tabulated.

### 8.2.2 Urinalysis

Urinalysis test results will be listed. All positive findings in the microscopic examination will be listed.

Observations outside the normal range will be flagged. The abnormal quantitative values will be flagged with 'L' for values below the lower limit of the laboratory's normal range, 'H' for values above the upper limit of the laboratory's normal range, or 'Ab' for abnormal qualitative test results. All original and unscheduled assessments will be listed.

### 8.3 Other Blood and Urine Samples

Details of the other blood and urine sample collections collected for pharmacogenomics, proteomics, genomics, metabolomics and lipidomics will be listed for each patient.

### 8.4 Vital Signs

The observed data for blood pressure (systolic and diastolic), heart rate (pulse), pulse oximetry, and body temperature will be listed by patient, and time point. Change from baseline values for blood pressure (systolic and diastolic), and heart rate (pulse) will be derived and listed. The baseline value to be used to derive change from baseline will be last assessment prior to first dose on Visit 2. The overall qualitative assessment for vital signs will be listed.

For systolic and diastolic blood pressure and heart rate, the observed values and change from baseline data will be summarized by treatment and time point. Table summaries will include descriptive statistics showing the number of observations (n), mean, SD, median, minimum, and maximum value.

### 8.5 12-Lead Safety ECG

Observed quantitative results for RR, PR, QRS, QT, QTcB (corrected QT according to Bazett), QTcF (corrected QT according to Fridericia) and heart rate will be listed for each patient. Change from baseline for QT, QTcB, QTcF will be derived and listed.

In the calculation of change from baseline, the baseline value for each period will be the last assessment prior to first dose on Visit 2.

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

The overall qualitative ECG assessment Abnormal NCS, Abnormal CS, and any comments will be listed for each patient.

For QT, QTcB, QTcF the observed and change from baseline data will be summarized by treatment and time point. Summaries will include tables of descriptive statistics showing the number of observations (n), mean, SD, median, minimum, and maximum value.

The number and percentage of patients having observed QT, QTcB, QTcF values that satisfy the following conditions will be summarized by treatment and time point:

- < 450 msec
- 450 < to < 480 msec
- $480 < \text{to} \le 500 \text{ msec}$
- > 500 msec

The number and percentage of patients having change from baseline QT, QTcB, QTcF values that satisfy the following conditions will be presented by treatment and time point:

- $\leq 0$  msec
- > 0 to < 30 msec
- $> 30 \text{ to} \le 60 \text{ msec}$
- > 60 msec

### 8.6 Physical Examination and Weight

All abnormal physical exam findings (pre and post-dose assessments) will be listed.

Patient weight collected pre and post dose will be listed.

### 8.7 Phone Call to Assess Safety

Results of this assessment will be listed for each patient and each visit.

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

### 9. **Reporting Output**

The following details the requirements and specifications for the presentation of the tables, figures and listings (TFLs) as set out in the TFL shells.

The tables, listings, figures and any non-descriptive statistical analysis will be produced using Unix SAS® Software (Version 9.2 or higher). The REPORT procedure will be used to produce all tables and listings; SAS/GRAPH will be used to produce all figures.

Tables, listings, and figures will be produced in the order that they appear in the textual sections of the plan.

All tables, listings, and graphs will be produced to landscape orientation using Courier New 8pt font and will be incorporated into a MS Word document as a (RTF) rich text file (margins: top, left, right, and bottom: 1 inch). Details are provided below.

- A separate RTF document will be created for each table, figure and listing individually.
- All TFLs will be produced in a landscape format, as far as is feasible.
- The standard font size and font type are "8 point", "Courier New" for all TFLs.
- Every page of each output will contain a footer indicating the date and time when the output was produced.
- Page numbering of tables and listings will use the format "Page X of Y". Page numbering for figures will be consecutive integers.
- The ordering of visits will be chronological
- Footnotes are left justified.

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

### 10. References

1. Murphy, L. B., et al. (2010). "Estimating medical costs attributable to osteoarthritis in the US population: comment on the article by Kotlarz et al." Arthritis and Rheumatism 62(8): 2566-2567; author reply 25672568.

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

### 11. Summary Tables

| TLF Number | Title | Topine<br>Item |
|---|---|---|
| Table 14.1.1 | Patient Disposition – All Enrolled Patients | Yes |
| Table 14.1.2.1 | Demographics - Continuous Variables, PPS Population | 103 |
| Table 14.1.2.2 | Demographics – Continuous Variables, mITT Population | |
| Table 14.1.3.1 | Demographics - Categorical Variables, PPS Population | |
| Table 14.1.3.2 | Demographics - Categorical Variables, mITT Population | |
| Table 14.1.4.1 | Prior Medications, PPS Population | |
| Table 14.1.4.2 | Prior Medications, mITT Population | |
| Table 14.1.5.1 | Concomitant Medications, PPS Population | |
| Table 14.1.5.2 | Concomitant, mITT Population | |
| Table 14.1.6 | Dose Administration - Number and Percentage of Patients Who<br>Received IMP by Visit, SAF Population | Yes |
| Table 14.1.7 | Dose Administration – Summary of Dosing Compliance, SAF Population | Yes |
| Pharmacoodyna | | |
| Table 14.2.1 | NRS Scores Observed and Change from Baseline Summary, mITT Population | |
| Table 14.2.2 | Number and Percentage of Patients by Category for Duration and Onset of Knee Pain at Baseline, mITT Population | |
| Table 14.2.3.1 | Statistical Analysis Primary Hypothesis - MIV-711 will Reduce Pain in Patients with Moderate Osteoarthritis - Assessments Using NRS Scores as Primary Endpoint, mITT Population | Yes |
| Table 14.2.3.2 | Statistical Analysis Primary Hypothesis - MIV-711 will Reduce Pain in Patients with Moderate Osteoarthritis - Assessments Using NRS Scores as Secondary Endpoints, mITT Population | |
| Table 14.2.3.3 | Statistical Analysis Primary Hypothesis - MIV-711 will Reduce Pain in Patients with Moderate Osteoarthritis - Assessments Using NRS Scores as Primary Endpoint, PPS Population | Yes |
| Table 14.2.3.4 | Statistical Analysis Primary Hypothesis - MIV-711 will Reduce Pain in Patients with Moderate Osteoarthritis - Assessments Using NRS Scores as Secondary Endpoints, PPS Population | |
| Table 14.2.4.1 | Imaging variables - MRI of Bone Area for the Target Knee Observed and Change from Baseline Summary, mITT Population | |
| Table 14.2.4.2 | Statistical Analysis - MRI of Bone Area for the Target Knee in Patients with Moderate Osteoarthritis, mITT Population | |
| Table 14.2.4.3 | Imaging variables - MRI of Cartilage Thickness for the Target Knee<br>Observed and Change from Baseline Summary, mITT Population | |
| Table 14.2.4.4 | Statistical Analysis - MRI of Cartilage Thickness for the Target Knee in Patients with Moderate Osteoarthritis, mITT Population | |
| Table 14.2.4.5 | Imaging variables - MRI of Total BML Volume for the Target Knee | |

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

| | Observed and Change from Baseline Summary, mITT Population | |
|---|---|---|
| Table 14.2.4.6 | Statistical Analysis - MRI of Total BML Volume for the Target Knee | |
| | in Patients with Moderate Osteoarthritis, mITT Population | |
| Table 14.2.4.7 | Other Imaging Variables MOAKS - Number and Percentage of | |
| | Subjects by Category and Treatment, mITT Population | |
| Table 14.2.4.8 | Other Imaging variables MOAKS - Observed and Change from | |
| | Baseline Summary, mITT Population | |
| Table 14.2.5 | Transformed ICOAP Scores Observed and Change from Baseline | |
| | Summary, mITT Population | |
| Table 14.2.6.1 | WOMAC Scores Observed and Change from Baseline Summary - Pain | |
| | Questions, mITT Population | |
| Table 14.2.6.2 | WOMAC Scores Observed and Change from Baseline Summary - | |
| | Stiffness Questions, mITT Population | |
| Table 14.2.6.3 | WOMAC Scores Observed and Change from Baseline Summary - | |
| | Difficulty Questions, mITT Population | |
| Table 14.2.7 | Number and Percentage of Patients with a Positive OARSI- | |
| | OMERACT Response, mITT Population | |
| Table 14.2.8 | Number and Percentage of Patients with Each Global Improvement | |
| | Score Response, mITT Population | |
| Table 14.2.9 | EQ-5D-5L Health Rating Score Response Observed and Change from | |
| | Baseline Summary, mITT Population | |
| Table 14.2.10.1 | E-Diary NRS Scores Observed and Change from Baseline Summary, | |
| | mITT Population, AM Response, mITT Population | |
| Table 14.2.10.2 | E-Diary NRS Scores Observed and Change from Baseline Summary, | |
| | mITT Population, PM Response, mITT Population | |
| Table 14.2.10.3 | E-Diary NRS Scores Observed and Change from Baseline Summary, | |
| | mITT Population, Overall Response, mITT Population | |
| Table 14.2.10.4 | Number and Percentage of Patients with E-Diary Pain Medication | |
| | Usage (Yes/No) Over Last 12 Hours, AM Response, mITT Population | |
| Table 14.2.10.5 | Number and Percentage of Patients with E-Diary Pain Medication | |
| | Usage (Yes/No) Over Last 12 Hours, PM Response, mITT Population | |
| Table 14.2.10.6 | Number and Percentage of Patients with E-Diary Pain Medication | |
| | Usage (Yes/No) Over Last 12 Hours, Overall Response, mITT | |
| | Population | |
| Table 14.2.10.7 | E-Diary Pain Medication Usage Number and Percentage of Patients | |
| | with each Reported Category, AM Response, mITT Population | |
| Table 14.2.10.8 | E-Diary Pain Medication Usage Number and Percentage of Patients | |
| | with each Reported Category, PM Response, mITT Population | |
| G 6 4 | | |
| Safety | C | X/ |
| Table 14.3.1.1 | Summary of Treatment Emergent Adverse Events, SAF Population | Yes |
| Table 14.3.1.2 | Number and Percentage of Patients with Treatment Emergent Adverse | Yes |
| | Events by System Organ Class, Preferred Term, and Treatment, SAF | |
| T-1-1- 142 12 | Population | V |
| Table 14.3.1.3 | Number and Percentage of Patients with Treatment Emergent | Yes |
| | Adverse Events 'Related to IMP' by System Organ Class, | <u> </u> |

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

| | Preferred Term, Severity, and Treatment, SAF Population |
|---|---|
| Table 14.3.1.4 | Number and Percentage of Patients with Treatment Emergent |
| | Adverse Events 'Not Related to IMP' by System Organ Class, |
| | Preferred Term, Severity, and Treatment, SAF Population |
| Table 14.3.1.5 | Number and Percentage of Patients with Serious Treatment Emergent |
| | Adverse Events by System Organ Class, Preferred Term, and |
| | Treatment, SAF Population |
| Table 14.3.1.6 | Number and Percentage of Patients with Treatment Emergent Adverse |
| | Events Leading to Discontinuation by System Organ Class, Preferred |
| | Term, and Treatment, SAF Population |
| Table 14.3.2.1 | Clinical Laboratory Chemistry Summary of Observed Values, SAF |
| | Population |
| Table 14.3.2.2 | Clinical Laboratory Hematology Summary of Observed Values, SAF |
| T 11 14 2 2 2 | Population Clinical Research C |
| Table 14.3.2.3 | Clinical Laboratory Chemistry – Shift From Baseline to Maximum |
| | Post-dose Value, SAF Population |
| Table 14.3.2.4 | Clinical Laboratory Chemistry – Shift From Baseline to Minimum |
| | Post-dose Value, SAF Population |
| Table 14.3.2.5 | Clinical Laboratory Hematology – Shift From Baseline to Maximum |
| | Post-dose Value, SAF Population |
| Table 14.3.2.6 | Clinical Laboratory Hematology – Shift From Baseline to Minimum |
| T. 11. 14.2.2 | Post-dose Value, SAF Population |
| Table 14.3.3 | Vital Signs Blood Pressure and Heart Rate Summary of Observed and |
| T. 11. 14.2.44 | Change from Baseline Values, SAF Population |
| Table 14.3.4.1 | 12 Lead ECG – Summary of Observed and Change from Baseline |
| T. 11. 14.2.4.2 | Values SAF Population |
| Table 14.3.4.2 | 12-Lead ECG – Categorical Summary of Observed Values, SAF |
| | Population |
| Table 14.3.4.3 | 12-Lead ECG – Categorical Summary of Change From Baseline, SAF |
| | Population |

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

### 12. **Figures**

| TLF Number | Title | Topline<br>Item |
|---|---|---|
| Figure 14.2.1 | Mean ± 95% CI Profiles of Observed NRS Scores | |
| Figure 14.2.2 | by Treatment, mITT Population Mean ± 95% CI Profiles of Change From Baseline | |
| rigule 14.2.2 | NRS Scores by Treatment, mITT Population | |
| Figure 14.2.3.1 | NRS Change From Baseline Scores (LSMean ± | |
| 1 iguic 14.2.3.1 | 95% CI) by Treatment and Time Point, mITT | |
| | Population | |
| Figure 14.2.3.2 | NRS Change From Baseline Scores (LSMean ± | |
| | 95% CI) by Treatment and Time Point, PPS | |
| | Population | |
| Figure 14.2.3.3 | NRS Change From Baseline (LSMean Difference ± | Yes |
| | 95% CI) Difference from Placebo by Treatment and | |
| | Time Point, mITT Population | |
| Figure 14.2.3.4 | NRS Change From Baseline (LSMean Difference ± | Yes |
| | 95% CI) Difference from Placebo by Treatment and | |
| | Time Point, PPS Population | |
| Figure 14.2.4.1 | MRI of Bone Area for the Target Knee - Mean | |
| | (SD) Change From Baseline Response over Time, | |
| | mITT Population | |
| Figure 14.2.4.2 | MRI of Bone Area for the Target Knee Change | |
| | From Baseline (LSMean Difference ± 95% CI) | |
| | Difference from Placebo by Treatment and Time | |
| | Point, mITT Population | |
| Figure 14.2.4.3 | MRI of Cartilage Thickness Change From Baseline | |
| | (LSMean Difference $\pm$ 95% CI) Difference from | |
| | Placebo by Treatment and Time Point, mITT | |
| | Population | |
| Figure 14.2.4.4 | MRI of Total BML Volume Change From Baseline | |
| | (LSMean Difference $\pm$ 95% CI) Difference from | |
| | Placebo by Treatment and Time Point, mITT | |
| | Population | |
| Figure 14.2.5 | ICOAP Mean Change From Baseline by Treatment | |
| 7: 112 (1 | and Time Point, mITT Population | |
| Figure 14.2.6.1 | WOMAC Pain Score Mean Change From Baseline | |
| 7: 112.62 | by Treatment and Time Point, mITT Population | |
| Figure 14.2.6.2 | WOMAC Stiffness Score Mean Change From | |
| | Baseline by Treatment and Time Point, mITT | |
| E: 140.63 | Population Classic Research | |
| Figure 14.2.6.3 | WOMAC Difficulty Score Mean Change From | |
| | Baseline by Treatment and Time Point, mITT | |
| | Population | |

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

| Figure 14.2.7 | |
|----------------|------------------------------------------------|
| | Scores (95% CI) by Treatment and Time |
| Figure 14.2.8 | Mean $\pm$ SD Profiles of Observed NRS E-Diary |
| | Scores by Treatment, mITT Population |
| Figure 14.2.9 | Mean ± SD Profiles of Change from Baseline NRS |
| | E-Diary Scores by Treatment, mITT Population |
| Figure 14.2.10 | Figures of Mean Response (95% CI) Over Time of |
| | Efficacy Biomarkers Serum CTX-I and Urinary |
| | CTX-II |

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

### 13. Listings

| | | Topline |
|---|---|---|
| TLF Number | Title | Item |
| Listing 16.2.1.1 | Patient Disposition | Yes |
| Listing 16.2.1.2 | Patients Excluded from Analysis Populations | Yes |
| Listing 16.2.1.3 | Enrolled Patients Who Did Not Meet All Eligibility Criteria | Yes |
| Listing 16.2.1.4 | Exclusion Tests | Yes |
| Listing 16.2.2.1 | Protocol Deviations | Yes |
| Listing 16.2.4.1 | Demographics | Yes |
| Listing 16.2.4.2 | Medical History | |
| Listing 16.2.5.1 | Prior and Concomitant Medications | Yes |
| Listing 16.2.5.2 | Dose Administration | Yes |
| Listing 16.2.5.3 | Dose Administration Compliance | |
| Listing 16.2.6.1 | Numerical Rating Scale of Knee Pain | |
| Listing 16.2.6.2 | Numerical Rating Scale of Knee Pain Change From Baseline | Yes |
| Listing 16.2.6.3 | Numerical Rating Scale of Knee Pain – Duration and Onset | Yes |
| Listing 16.2.6.4 | Imaging Results - MRI of Bone Area for the Target Knee | |
| Listing 16.2.6.5 | Imaging Results - MRI of Cartilage Thickness for the Target Knee | |
| Listing 16.2.6.6 | Other Secondary Imaging Variables – MOAKS | |
| Listing 16.2.6.7 | Other Secondary Imaging Variables Change From Baseline – | |
| | MOAKS | |
| Listing 16.2.6.8 | Other Secondary Imaging Variables – Imorphics | |
| Listing 16.2.6.9 | Other Secondary Imaging Variables Change From Baseline – | |
| | Imorphics | |
| Listing 16.2.6.10 | Observed Raw ICOAP Scores | |
| Listing 16.2.6.11 | Transformed ICOAP Scores | |
| Listing 16.2.6.12 | Western Ontario and McMaster Index (WOMAC) - Pain Questions | |
| Listing 16.2.6.13 | Western Ontario and McMaster Index (WOMAC) - Stiffness | |
| | Questions | |
| Listing 16.2.6.14 | Western Ontario and McMaster Index (WOMAC) - Difficulty | |
| | Questions | |
| Listing 16.2.6.15 | Western Ontario and McMaster Index (WOMAC) Change From | |
| | Baseline - Pain Questions | |
| Listing 16.2.6.16 | Western Ontario and McMaster Index (WOMAC) Change From | |
| | Baseline - Stiffness Questions | |
| Listing 16.2.6.17 | Western Ontario and McMaster Index (WOMAC) Change From | |
| | Baseline - Difficulty Questions | |
| Listing 16.2.6.18 | OARSI-OMERACT Responder Index Derived Scores out of 100 | |
| Listing 16.2.6.19 | OARSI-OMERACT Responder Index | |
| | Change from Baseline and Percentage Change from Baseline | |
| | Scores | |
| Listing 16.2.6.20 | Global Improvements | |
| Listing 16.2.6.21 | Quality of Life Patient Reported Outcomes - EQ-5D-5L | |

Medivir Final 1.0 Protocol: MIV-711-201 22 June 2017

| Listing 16.2.6.22 | Quality of Life Patient Reported Outcomes Change from Baseline |
|---|---|
| | Scores - EQ-5D-5L |
| Listing 16.2.6.23 | Brief Medication Questionnaire |
| Listing 16.2.6.24 | E-Diary |
| Listing 16.2.6.25 | Efficacy Biomarkers from Serum and Urine Samples |
| Listing 16.2.6.26 | Time-Integrated Concentrations (TIC) and Their Z-scores |
| | for Efficacy Biomarkers from Serum and Urine Samples |
| Listing 16.2.7.1 | Adverse Events |
| Listing 16.2.7.2 | Serious Adverse Events |
| Listing 16.2.7.3 | Adverse Events Leading to Discontinuation |
| Listing 16.2.8.1 | Clinical Laboratory Chemistry – Observed Values |
| Listing 16.2.8.2 | Clinical Laboratory Hematology – Observed Values |
| Listing 16.2.8.3 | Clinical Laboratory Urinalysis – Observed Values |
| Listing 16.2.8.4 | Clinical Laboratory Urinalysis – Positive Microscopic Findings |
| Listing 16.2.8.5 | Vital Signs Observed Values |
| Listing 16.2.8.6 | Vital Signs Change from Baseline |
| Listing 16.2.8.7 | Vital Signs Overall Qualitative Results Abnormal Assessments |
| Listing 16.2.8.8 | 12 Lead ECG Quantitative Findings |
| Listing 16.2.8.9 | 12 Lead ECG Change From Baseline |
| Listing 16.2.8.10 | 12 Lead ECG Overall Qualitative Assessment |
| Listing 16.2.8.11 | Physical Examination Abnormal Findings |
| Listing 16.2.8.12 | Patient Weight |
| Listing 16.2.8.13 | Phone Call to Assess Safety |

Medivir
Protocol: 012-01

22 June 2017

### 14. Table Shells

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Page X of Y

Medivir

Protocol Number: MIV-711-201

Table 14.1.1
Patient Disposition
All Enrolled Patients

| | | Treatment | | |
|---|---|---|---|---|
| | Placebo<br>N = x | 100 mg<br>MIV-711<br>N = x | 200 mg<br>MIV-711<br>N = x | Overall<br>N = x |
| Number Patients Enrolled | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Completed Study | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Discontinued from Study | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Number Patients in ITT Population | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Number Patients in mITT Population | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Number Patients in PPS Population | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Number Patients in SAF Population | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Reason for Discontinuation | | | | |
| Adverse Event | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Protocol Deviation | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Consent Withdrawn | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Lost to Follow-Up | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Death | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Other | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |

Medivir

Protocol: MIV-711-201

22 June 2017

Final 1.0

Medivir

Protocol Number: MIV-711-201

Page X of Y

Table 14.1.2.1

Demographics - Continuous Variables

PPS Population

| | | | Treatment | | |
|---|---|---|---|---|---|
| | Statistic | Placebo<br>N = x | 100 mg<br>MIV-711<br>N = x | 200 mg<br>MIV-711<br>N = x | Overall<br>N = x |
| | n | nn | nn | nn | nn |
| | Mean | XX.X | XX.X | XX.X | XX.X |
| Age | SD | XX.XX | XX.XX | XX.XX | XX.XX |
| (years) | Median | XX.X | XX.X | XX.X | XX.X |
| | Min | XX | XX | XX | XX |
| | Max | XX | XX | XX | XX |
| | n | nn | nn | nn | nn |
| | Mean | XX.X | XX.X | XX.X | XX.X |
| Height | SD | XX.XX | XX.XX | XX.XX | XX.XX |
| (cm) | Median | XX.X | XX.X | XX.X | XX.X |
| (01) | Min | XX | XX | XX | XX |
| | Max | XX | XX | XX | xx |
| | _ | | | | |
| | n | nn | nn | nn | nn |
| Total subst | Mean | XX.X | XX.X | XX.X | XX.X |
| Weight | SD | XX.XX | XX.XX | XX.XX | XX.XX |
| (kg) | Median | XX.X | XX.X | XX.X | XX.X |
| | Min | XX | XX | XX | XX |
| | Max | XX | XX | XX | XX |
| | n | nn | nn | nn | nn |
| | Mean | XX.X | XX.X | XX.X | XX.X |
| BMI | SD | XX.XX | XX.XX | XX.XX | XX.XX |
| (kg/m^2) | Median | XX.X | XX.X | XX.X | XX.X |
| | Min | XX | XX | XX | XX |
| | Max | XX | XX | XX | XX |

Programming note: table will be created for mITT population: Table 14.1.2.2 Demographics - Continuous Variables, mITT Population

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Page X of Y

Medivir

Protocol Number: MIV-711-201

Table 14.1.3.1

Demographics - Categorical Variables

PPS Population

Treatment

| | Placebo N = x | | | -<br>Overall |
|---|---|---|---|---|
| | | N = x | $ MIV-711 \\ N = x $ | N = x |
| Ethnicity | | | | |
| Hispanic/Latino | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Non-Hispanic/Latino | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Race | | | | |
| White | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| American Indian/Alaska Native | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Asian | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Native Hawaiian or other Pacific Islander | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Black/African American | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Other | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Gender | | | | |
| Female | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Male | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |

Programming note: table will be created for mITT population: Table 14.1.3.2 Demographics - Categorical Variables, mITT Population

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Page X of Y

Medivir

Protocol Number: MIV-711-201

Table 14.1.4.1
Prior Medications
PPS Population

| | | • | | |
|---|---|---|---|---|
| ATC Classification | Placebo<br>N = x | 100 mg<br>MIV-711<br>N = x | 200 mg<br>MIV-711<br>N = x | Overall<br>N = x |
| | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |

Programming note: table will be created for mITT population: Table 14.1.4.2 Prior Medications, mITT Population

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Table 14.1.5.1 Concomitant Medications PPS Population

| | Treatment | | | |
|---|---|---|---|---|
| ATC Classification | Placebo<br>N = x | 100 mg<br>MIV-711<br>N = x | 200 mg<br>MIV-711<br>N = x | Overall<br>N = x |
| | nn (nn.n%)<br>nn (nn.n%) | nn (nn.n%)<br>nn (nn.n%) | nn (nn.n%)<br>nn (nn.n%) | nn (nn.n%)<br>nn (nn.n%) |

Programming note: table will be created for mITT population: Table 14.1.5.2 Concomitant Medications, mITT Population

Medivir

Final 1.0 22 June 2017 Protocol: MIV-711-201

Page X of Y Medivir Protocol Number: MIV-711-201

Table 14.1.6 Dose Administration - Number and Percentage of Patients Who Received IMP by Visit

| | | Treatment | | |
|---|---|---|---|---|
| Visit | Placebo<br>N = x | 100 mg<br>MIV-711 | 200 mg<br>MIV-711 | Overall |
| | | N = x | N = X | N = x |
| VISIT 2 BASELINE DAY 1 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| VISIT 5 WEEK 8 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| VISIT 6 WEEK 14 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |

SAF Population

Etc...

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Table 14.1.7
Summary of Dosing Compliance
SAF Population

| | | | | - | |
|---|---|---|---|---|---|
| | Statistic | Placebo<br>N = x | 100 mg<br>MIV-711<br>N = x | 200 mg<br>MIV-711<br>N = x | Overall<br>N = x |
| | n | nn | nn | nn | nn |
| Planned | Mean | XX.X | XX.X | XX.X | XX.X |
| Number of | SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Days IMP | Median | XX.X | XX.X | XX.X | XX.X |
| exposure | Min | XX | XX | XX | XX |
| | Max | XX | XX | XX | XX |
| Actual<br>Number of<br>Capsules<br>used | n<br>Mean<br>SD<br>Median<br>Min<br>Max | nn<br>xx.x<br>xx.xx<br>xx.x<br>xx.x | nn<br>xx.x<br>xx.xx<br>xx.x<br>xx.x | nn<br>xx.x<br>xx.xx<br>xx.x<br>xx.x | nn<br>xx.x<br>xx.xx<br>xx.x<br>xx.x |
| IMP<br>Compliance<br>(%) | n<br>Mean<br>SD<br>Median<br>Min<br>Max | nn<br>xx.x<br>xx.xx<br>xx.x<br>xx.x | nn<br>xx.x<br>xx.xx<br>xx.x<br>xx.x | nn<br>xx.x<br>xx.xx<br>xx.x<br>xx | nn<br>xx.x<br>xx.xx<br>xx.x<br>xx |

The 'actual number of capsules used' was derived as the 'number of capsules dispensed' minus the 'number of capsules returned'.

'Planned number of capsules' is the number of days of per protocol dosing from V2 (first dose) to V8 (last dose), since each patient is to receive 1 capsule of dosing per day of dose administration.

IMP compliance: (actual number of capsules used / planned number of capsules administered) x 100%

Medivir

Protocol: MIV-711-201

22 June 2017

Page X of Y

Final 1.0

Medivir

Protocol Number: MIV-711-201

Table 14.2.1

NRS Scores Observed and Change from Baseline Summary

mITT Population

Parameter = How Active the target knee arthritis has been

| | | | | Treati | ment | | |
|---|---|---|---|---|---|---|---|
| | | Place | ebo | 100<br>MIV- | _ | 200 mg<br>MIV-711 | |
| | | Observed | Change | Observed | Change | Observed | Change |
| Visit | Statistic | N = x | N = x | N = x | N = x | N = x | N = x |
| | n | nn | | nn | | nn | |
| | Mean | XX.X | | XX.X | | XX.X | |
| VISIT 2 | SD | XX.XX | | XX.XX | | XX.XX | |
| Baseline | Median | XX.X | | XX.X | | XX.X | |
| | Min | XX | | XX | | XX | |
| | Max | XX | | xx | | xx | |
| | n | nn | nn | nn | nn | nn | nn |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| VISIT 5 | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| WEEK 8 | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min | XX | XX | XX | XX | XX | XX |
| | Max | XX | XX | XX | XX | XX | XX |
| | n | nn | nn | nn | nn | nn | nn |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| VISIT 6 | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | xx.xx |
| WEEK 14 | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min | XX | XX | XX | XX | XX | XX |
| | Max | XX | XX | XX | XX | XX | XX |
| Et.c | | | | | | | |

Etc...

Programming note: table will include summaries for following other NRS scores:

- Primary endpoint: Amount of pain severity in the target knee last week (SDTM: Overall pain severity in target knee
- Global Assessment Score: How active has the target knee arthritis has been in the past week (SDTM: How active was target knee arthritis)
- Satisfaction with target knee function (SDTM: How satisfied are you with target knee function)
- Worst pain severity in target knee (SDTM: Worst pain severity in target knee)
- Overall pain severity in other knee (SDTM: Overall pain severity in other knee)

Medivir
Protocol: MIV-711-201
22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Table 14.2.2

Number and Percentage of Patients by Category for Duration and Onset of Knee Pain at Baseline

mITT Population

Parameter = Duration of Knee Pain Past 12 Months

| | Treatment | | |
|---|---|---|---|
| Category | Placebo<br>N = x | 100 mg<br>MIV-711<br>N = x | 200 mg<br>MIV-711<br>N = x |
| | nn (nn.n%)<br>nn (nn.n%)<br>nn (nn.n%) | nn (nn.n%)<br>nn (nn.n%)<br>nn (nn.n%) | nn (nn.n%)<br>nn (nn.n%)<br>nn (nn.n%) |

Etc...

Programming note: table will include summaries for:

- Duration of Knee Pain Past 12 Months
- Onset of Knee Pain

Medivir

Protocol: MIV-711-201 22 June 2017

Medivir Page X of Y

Protocol Number: MIV-711-201

Table 14.2.3.1

Statistical Analysis Primary Hypothesis - MIV-711 will Reduce Pain in Patients with Moderate Osteoarthritis
Assessments Using NRS Scores as Primary Endpoint
mITT Population

| | | | | | | Diffe | rence From |
|---|---|---|---|---|---|---|---|
| | | | | Change From | n Baseline NRS | P | lacebo |
| Question | Treatment | Week | | LS | | LS Mean | |
| | | | N | Mean | 95% CI | Difference | 95% CI |
| | Placebo | 8 | nn | XX.XX | (x.xx, x.xx) | | |
| | | 14 | nn | XX.XX | (x.xx, x.xx) | | |
| | | 26 | nn | XX.XX | (xx.x, xx.x) | | |
| | | 30 | nn | XX.XX | (x.xx, x.xx) | | |
| NRS question | 100 mg MIV-711 | 8 | nn | XX.XX | (x.xx, x.xx) | XX.XX | (x.xx, x.xx) |
| 1: Pain severity in | | 14 | nn | XX.XX | (x.xx, x.xx) | XX.XX | (x.xx, x.xx) |
| target knee | | 26 | nn | XX.XX | (xx.x, xx.x) | XX.XX | (x.xx, x.xx) |
| [last week] | | 30 | nn | XX.XX | (x.xx, x.xx) | xx.xx | (xx.x, xx.x) |
| | 200 mg MIV-711 | 8 | nn | XX.XX | (x.xx, x.xx) | XX.XX | (x.xx, x.xx) |
| | | 14 | nn | XX.XX | (x.xx, x.xx) | XX.XX | (x.xx, x.xx) |
| | | 26 | nn | XX.XX | (xx.x, xx.x) | xx.xx | (x.xx, x.xx) |
| | | 30 | nn | XX.XX | (x.xx, x.xx) | XX.XX | (xx.x, xx.x) |

LS Mean = least squares mean, N denotes the number of Patients for each level of treatment used to estimate the LS means. Programming notes:

Low pain scores are associated with a positive outcome (effect of drug).

For positive study expect large (negative changes from week 26) decreases from baseline by the time treatment reaches week 26.

Final 1.0

Medivir

Final 1.0 Protocol: MIV-711-201 22 June 2017

Medivir Page X of Y

Protocol Number: MIV-711-201

Table 14.2.3.2

Statistical Analysis Primary Hypothesis - MIV-711 will Reduce Pain in Patients with Moderate Osteoarthritis Assessments Using NRS Scores as Secondary Endpoints mITT Population

| | | | | | | | rence From |
|---|---|---|---|---|---|---|---|
| | | | | Change From | n Baseline NRS | P | lacebo |
| Question | Treatment | Week | | LS | | LS Mean | |
| | | | N | Mean | 95% CI | Difference | 95% CI |
| | Placebo | 8 | nn | XX.XX | (x.xx, x.xx) | | |
| | | 14 | nn | XX.XX | (x.xx, x.xx) | | |
| | | 26 | nn | XX.XX | (xx.x, xx.x) | | |
| | | 30 | nn | XX.XX | (x.xx, x.xx) | | |
| Global | 100 mg MIV-711 | 8 | nn | XX.XX | (x.xx, x.xx) | xx.xx | (x.xx, x.xx) |
| Assessment<br>Score: How | | 14 | nn | XX.XX | (x.xx, x.xx) | XX.XX | (x.xx, x.xx) |
| active was | | 26 | nn | XX.XX | (xx.x, xx.x) | XX.XX | (x.xx, x.xx) |
| target knee | | 30 | nn | XX.XX | (x.xx, x.xx) | xx.xx | (xx.x, xx.x) |
| arthritis | | | | | | | |
| | 200 mg MIV-711 | 8 | nn | XX.XX | (x.xx, x.xx) | xx.xx | (x.xx, x.xx) |
| | | 14 | nn | XX.XX | (x.xx, x.xx) | XX.XX | (x.xx, x.xx) |
| | | 26 | nn | XX.XX | (xx.x, xx.x) | xx.xx | (x.xx, x.xx) |
| | | 30 | nn | xx.xx | (x.xx, x.xx) | xx.xx | (xx.x, xx.x) |

LS Mean = least squares mean, N denotes the number of Patients for each level of treatment used to estimate the LS means. Programming notes:

Low pain scores are associated with a positive outcome (effect of drug).

For positive study expect large (negative changes from week 26) decreases from baseline by the time treatment reaches week 26.

Table will be expanded to include the analysis of the following NRS scores:

- Global Assessment Score: How active has the target knee arthritis has been in the past week (SDTM: How active was target knee arthritis)
- Satisfaction with target knee function (SDTM:How satisfied are you with target knee function)
- Worst pain severity in target knee (SDTM: Worst pain severity in target knee)
- Overall pain severity in other knee (SDTM: Overall pain severity in other knee)

Medivir

Final 1.0 Protocol: MIV-711-201 22 June 2017

Medivir Page X of Y

Protocol Number: MIV-711-201

Table 14.2.3.3 Statistical Analysis Primary Hypothesis - MIV-711 will Reduce Pain in Patients with Moderate Osteoarthritis Assessments Using NRS Scores as Primary Endpoint PPS Population

| | | | | | | | rence From |
|---|---|---|---|---|---|---|---|
| | | | | Change From | n Baseline NRS | P | lacebo |
| Question | Treatment | Week | | LS | | LS Mean | |
| | | | N | Mean | 95% CI | Difference | 95% CI |
| | Placebo | 8 | nn | XX.XX | (x.xx, x.xx) | | |
| | | 14 | nn | XX.XX | (x.xx, x.xx) | | |
| | | 26 | nn | XX.XX | (xx.x, xx.x) | | |
| | | 30 | nn | XX.XX | (x.xx, x.xx) | | |
| NRS question | 100 mg MIV-711 | 8 | nn | XX.XX | (x.xx, x.xx) | xx.xx | (x.xx, x.xx) |
| 1: Pain severity in | | 14 | nn | XX.XX | (x.xx, x.xx) | XX.XX | (x.xx, x.xx) |
| target knee | | 26 | nn | XX.XX | (xx.x, xx.x) | XX.XX | (x.xx, x.xx) |
| [last week] | | 30 | nn | XX.XX | (x.xx, x.xx) | xx.xx | (xx.x, xx.x) |
| | 200 mg MIV-711 | 8 | nn | XX.XX | (x.xx, x.xx) | xx.xx | (x.xx, x.xx) |
| | | 14 | nn | XX.XX | (x.xx, x.xx) | xx.xx | (x.xx, x.xx) |
| | | 26 | nn | XX.XX | (xx.x, xx.x) | xx.xx | (x.xx, x.xx) |
| | | 30 | nn | XX.XX | (x.xx, x.xx) | xx.xx | (xx.x, xx.x) |

LS Mean = least squares mean, N denotes the number of Patients for each level of treatment used to estimate the LS means. Programming notes:

Low pain scores are associated with a positive outcome (effect of drug).

For positive study expect large (negative changes from week 26) decreases from baseline by the time treatment reaches week 26.

Medivir

Final 1.0 Protocol: MIV-711-201 22 June 2017

Medivir Page X of Y

Protocol Number: MIV-711-201

Table 14.2.3.4

Statistical Analysis Primary Hypothesis - MIV-711 will Reduce Pain in Patients with Moderate Osteoarthritis Assessments Using NRS Scores as Secondary Endpoints PPS Population

| | | | | | | | rence From |
|---|---|---|---|---|---|---|---|
| | | | | Change From | n Baseline NRS | PI | .acebo |
| Question | Treatment | Week | | LS | | LS Mean | |
| | | | N | Mean | 95% CI | Difference | 95% CI |
| | Placebo | 8 | nn | XX.XX | (x.xx, x.xx) | | |
| | | 14 | nn | XX.XX | (x.xx, x.xx) | | |
| | | 26 | nn | XX.XX | (xx.x, xx.x) | | |
| | | 30 | nn | XX.XX | (x.xx, x.xx) | | |
| Global | 100 mg MIV-711 | 8 | nn | XX.XX | (x.xx, x.xx) | XX.XX | (x.xx, x.xx) |
| Assessment<br>Score: How | | 14 | nn | XX.XX | (x.xx, x.xx) | XX.XX | (x.xx, x.xx) |
| active was | | 26 | nn | XX.XX | (xx.x, xx.x) | XX.XX | (x.xx, x.xx) |
| target knee | | 30 | nn | XX.XX | (x.xx, x.xx) | XX.XX | (xx.x, xx.x) |
| arthritis | | | | | | | |
| | 200 mg MIV-711 | 8 | nn | XX.XX | (x.xx, x.xx) | xx.xx | (x.xx, x.xx) |
| | | 14 | nn | XX.XX | (x.xx, x.xx) | xx.xx | (x.xx, x.xx) |
| | | 26 | nn | XX.XX | (xx.x, xx.x) | XX.XX | (x.xx, x.xx) |
| | | 30 | nn | XX.XX | (x.xx, x.xx) | XX.XX | (xx.x, xx.x) |

LS Mean = least squares mean, N denotes the number of Patients for each level of treatment used to estimate the LS means. Programming notes:

Low pain scores are associated with a positive outcome (effect of drug).

For positive study expect large (negative changes from week 26) decreases from baseline by the time treatment reaches week 26.

Table will be expanded to include the analysis of the following NRS scores:

- Global Assessment Score: How active has the target knee arthritis has been in the past week (SDTM: How active was target knee arthritis)
- Satisfaction with target knee function (SDTM:How satisfied are you with target knee function)
- Worst pain severity in target knee (SDTM: Worst pain severity in target knee)
- Overall pain severity in other knee (SDTM: Overall pain severity in other knee)

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Page X of Y

Medivir

Protocol Number: MIV-711-201

Table 14.2.4.1

Imaging variables - MRI of Bone Area for the Target Knee Observed and Change from Baseline Summary mITT Population

| | | | | Treatr | ment | | |
|---|---|---|---|---|---|---|---|
| | | Placebo | | 100<br>MIV- | _ | 200 mg<br>MIV-711 | |
| | | Observed | Change | Observed | Change | Observed | Change |
| Visit | Statistic | N = x | N = x | N = x | N = x | N = x | N = x |
| | n | nn | | nn | | nn | |
| | Mean | XX.X | | XX.X | | XX.X | |
| VISIT 2 | SD | XX.XX | | XX.XX | | XX.XX | |
| Baseline | Median | XX.X | | XX.X | | XX.X | |
| | Min | XX | | XX | | XX | |
| | Max | XX | | XX | | XX | |
| | n | nn | nn | nn | nn | nn | nn |
| | Mean | xx.x | xx.x | XX.X | xx.x | XX.X | XX.X |
| VISIT 8 | SD | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx |
| WEEK 26 | Median | xx.x | xx.x | XX.X | xx.x | XX.X | xx.x |
| | Min | XX | XX | XX | XX | XX | XX |
| | Max | XX | XX | XX | XX | XX | XX |

Programming note: source data obtained from MF\_TAB: Area of bone in the medial femur region, MF

Medivir
Protocol: MIV-711-201
22 June 2017

Medivir Page X of Y

Protocol Number: MIV-711-201

| | Change From Baseline NRS Difference From (Visit 8 Week 26) Placebo | | | | | |
|---|---|---|---|---|---|---|
| Question | Treatment | N | LS<br>Mean | 95% CI | LS Mean<br>Difference | 95% CI |
| | Placebo | nn | XX.XX | (x.xx, x.xx) | | |
| MRI of Bone<br>Area | 100 mg MIV-711 | nn | xx.xx | (x.xx, x.xx) | xx.xx | (x.xx, x.xx) |
| | 200 mg MIV-711 | nn | xx.xx | (x.xx, x.xx) | xx.xx | (x.xx, x.xx) |

LS Mean = least squares mean, N denotes the number of Patients for each level of treatment used to estimate the LS means. Programming notes:

Programming note: source data obtained from MF TAB: Area of bone in the medial femur region, MF

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Page X of Y

Medivir

Protocol Number: MIV-711-201

Table 14.2.4.3

Imaging variables - MRI of Cartilage Thickness for the Target Knee Observed and Change from Baseline Summary mITT Population

Parameter = Femur Region

| | | Treatment | | | | | |
|---|---|---|---|---|---|---|---|
| | | Placebo | | 100 mg<br>MIV-711 | | 200 mg<br>MIV-711 | |
| | | Observed | Change | Observed | Change | Observed | Change |
| Visit | Statistic | N = x | N = x | N = x | N = x | N = x | N = x |
| | n | nn | | nn | | nn | |
| | Mean | XX.X | | XX.X | | XX.X | |
| VISIT 2 | SD | XX.XX | | XX.XX | | XX.XX | |
| Baseline | Median | XX.X | | XX.X | | XX.X | |
| | Min | XX | | XX | | XX | |
| | Max | XX | | XX | | XX | |
| | n | nn | nn | nn | nn | nn | nn |
| | Mean | XX.X | xx.x | XX.X | xx.x | XX.X | xx.x |
| VISIT 8 | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| WEEK 26 | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min | XX | XX | XX | XX | XX | XX |
| | Max | XX | XX | XX | XX | XX | XX |

Programming note: source data obtained from:

- CM\_FEMUR\_THCTAB: Average thickness of cartilage in the central medial femur region
- CM\_TIBIA\_THCTAB: Average thickness of cartilage in the central medial tibia region

Medivir
Protocol: MIV-711-201
22 June 2017

Medivir Page X of Y

Protocol Number: MIV-711-201

| | | | Change From Baseline NRS<br>(Visit 8 Week 26) | | Difference From<br>Placebo | |
|---|---|---|---|---|---|---|
| Parameter | Treatment | | LS | | LS Mean | |
| | | N | Mean | 95% CI | Difference | 95% CI |
| | Placebo | nn | XX.XX | (x.xx, x.xx) | | |
| Femur Region | | | | | | |
| | 100 mg MIV-711 | nn | XX.XX | (x.xx, x.xx) | XX.XX | (x.xx, x.xx) |
| | 200 mg MIV-711 | nn | XX.XX | (x.xx, x.xx) | XX.XX | (x.xx, x.xx) |
| Etc | | | | | | |

LS Mean = least squares mean, N denotes the number of Patients for each level of treatment used to estimate the LS means. Programming notes:

Programming note: source data obtained from:

- CM FEMUR THCTAB: Average thickness of cartilage in the central medial femur region
- CM TIBIA THCTAB: Average thickness of cartilage in the central medial tibia region

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Page X of Y

Medivir

Protocol Number: MIV-711-201

Table 14.2.4.5

 $\hbox{Imaging variables - MRI of Total BML Volume for the Target Knee Observed and Change from Baseline Summary \\ \hbox{mITT Population}$ 

Parameter = Femur Region

| | | Treatment | | | | | |
|---|---|---|---|---|---|---|---|
| | | Placebo | | 100 mg<br>MIV-711 | | 200 mg<br>MIV-711 | |
| | | Observed | Change | Observed | Change | Observed | Change |
| Visit | Statistic | N = x | N = x | N = x | N = x | N = x | N = x |
| | n | nn | | nn | | nn | |
| | Mean | XX.X | | XX.X | | XX.X | |
| VISIT 2 | SD | XX.XX | | XX.XX | | XX.XX | |
| Baseline | Median | XX.X | | XX.X | | XX.X | |
| | Min | XX | | XX | | XX | |
| | Max | XX | | XX | | XX | |
| | n | nn | nn | nn | nn | nn | nn |
| | Mean | XX.X | xx.x | XX.X | xx.x | XX.X | xx.x |
| VISIT 8 | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| WEEK 26 | Median | XX.X | xx.x | XX.X | xx.x | XX.X | XX.X |
| | Min | XX | XX | XX | XX | XX | XX |
| | Max | XX | XX | XX | XX | XX | xx |

Programming note: source data obtained from: TOTAL\_BML\_VOLUME

Medivir
Protocol: MIV-711-201
22 June 2017

Medivir Page X of Y

Protocol Number: MIV-711-201

| | | | Change From Baseline NRS<br>(Visit 8 Week 26) | | Difference From<br>Placebo | |
|---|---|---|---|---|---|---|
| Parameter | Treatment | | LS | | LS Mean | |
| | | N | Mean | 95% CI | Difference | 95% CI |
| | Placebo | nn | XX.XX | (x.xx, x.xx) | | |
| Femur Region | | | | | | |
| | 100 mg MIV-711 | nn | XX.XX | (x.xx, x.xx) | XX.XX | (x.xx, x.xx) |
| | 200 mg MIV-711 | nn | XX.XX | (x.xx, x.xx) | XX.XX | (x.xx, x.xx) |
| Etc | | | | | | |

LS Mean = least squares mean, N denotes the number of Patients for each level of treatment used to estimate the LS means. Programming notes:

Programming note: source data obtained from: TOTAL BML VOLUME

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Table 14.2.4.7
Other Imaging variables MOAKS and Imorphics
Number and Percentage of Subjects by Category and Treatment
mITT Population

| | - | Treatment | | |
|---|---|---|---|---|
| | | Placebo | 100 mg<br>MIV-711 | 200 mg<br>MIV-711 |
| | Catgeory | N = x | N = x | N = x |
| Size of BML | None | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | <33% | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | 33-66% | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | >66% | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Not Evaluable | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Percentage that is BML | None | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | <33% | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | 33-66% | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | >66% | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Not Evaluable | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Etc | Etc | | | |

Programming note: table will include summaries for the MOAKS and Imorphics imaging variables collected using a categorical response
Medivir

Protocol: MIV-711-201

Medivir

Protocol Number: MIV-711-201

Table 14.2.4.8

Other Imaging variables MOAKS and Imorphics Observed and Change from Baseline Summary  $$\operatorname{\mathtt{mITT}}$$  Population

Parameter = Number of Bone Marrow Lesions

| | | | Treatment | | | | |
|---|---|---|---|---|---|---|---|
| | | Place | Placebo | | 100 mg<br>MIV-711 | | 200 mg<br>MIV-711 |
| | | Observed | Change | Observed | Change | Observed | Change |
| Visit | Statistic | N = x | N = x | N = x | N = x | N = x | N = x |
| | n | nn | | nn | | nn | |
| | Mean | XX.X | | XX.X | | XX.X | |
| VISIT 2 | SD | XX.XX | | XX.XX | | XX.XX | |
| Baseline | Median | XX.X | | XX.X | | XX.X | |
| | Min | XX | | XX | | XX | |
| | Max | XX | | XX | | XX | |
| | n | nn | nn | nn | nn | nn | nn |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| VISIT 8 | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| WEEK 26 | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min | XX | XX | XX | XX | XX | XX |
| | Max | XX | XX | XX | XX | XX | XX |

Programming note: table will include summaries for the other MOAKS and Imorphics variables collected using a quantitative response

Final 1.0

Page X of Y

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Page X of Y

Medivir

Protocol Number: MIV-711-201

Parameter = Constant Pain

| | | | | Treatr | ment | | |
|---|---|---|---|---|---|---|---|
| | | Placebo | | | 100 mg<br>MIV-711 | | 200 mg<br>MIV-711 |
| | | Observed | Change | Observed | Change | Observed | Change |
| Visit | Statistic | N = x | N = x | N = x | N = x | N = x | N = x |
| | n | nn | | nn | | nn | |
| | Mean | xx.x | | XX.X | | XX.X | |
| VISIT 2 | SD | XX.XX | | xx.xx | | xx.xx | |
| Baseline | Median | xx.x | | XX.X | | XX.X | |
| | Min | XX | | XX | | XX | |
| | Max | XX | | XX | | XX | |
| | n | nn | nn | nn | nn | nn | nn |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| VISIT 5 | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| WEEK 8 | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min | XX | XX | XX | XX | XX | XX |
| | Max | XX | XX | xx | XX | xx | XX |
| | n | nn | nn | nn | nn | nn | nn |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| VISIT 6 | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| WEEK 14 | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min | XX | XX | XX | XX | XX | XX |
| | Max | XX | XX | XX | XX | XX | XX |
| Etc | | | | | | | |

Programming note: table will include summaries for following transformed ICOAP scores: Constant Pain, Intermittent Pain, and Total Pain.

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Page X of Y

Medivir

Protocol Number: MIV-711-201

Table 14.2.6.1

WOMAC Scores Observed and Change from Baseline Summary - Pain Questions mITT Population

Parameter = Walking on flat surface

| | | | | Treatr | ment | | |
|---|---|---|---|---|---|---|---|
| | | Placebo | | | 100 mg<br>MIV-711 | | 200 mg<br>MIV-711 |
| | | Observed | Change | Observed | Change | Observed | Change |
| TT - 1 h | Quantitatia | | <u> </u> | | <u> </u> | | , |
| Visit | Statistic | N = x | N = x | N = x | N = x | N = x | N = x |
| | n<br>Mana | nn | | nn | | nn | |
| VISIT 2 | Mean<br>SD | XX.X | | XX.X | | XX.X | |
| Baseline | Median | xx.xx<br>xx.x | | XX.XX<br>XX.X | | XX.XX<br>XX.X | |
| Daserine | Min | | | | | | |
| | Max | XX<br>XX | | XX | | XX | |
| | Max | XX | | XX | | XX | |
| | n | nn | nn | nn | nn | nn | nn |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| VISIT 5 | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| WEEK 8 | Median | XX.X | xx.x | XX.X | XX.X | XX.X | XX.X |
| | Min | XX | XX | XX | XX | XX | XX |
| | Max | XX | XX | XX | XX | XX | XX |
| | n | nn | nn | nn | nn | nn | nn |
| | Mean | xx.x | xx.x | XX.X | xx.x | XX.X | XX.X |
| VISIT 6 | SD | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | XX.XX |
| WEEK 14 | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min | XX | XX | XX | XX | XX | XX |
| | Max | XX | XX | XX | XX | XX | XX |
| Etc | | | | | | | |

Programming note: table will be expanded to include all WOMAC Pain questions

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Page X of Y

Medivir

Protocol Number: MIV-711-201

Parameter = Stiffness after First Woke Up in Morning

| | | | | Treati | ment | | |
|---|---|---|---|---|---|---|---|
| | | Place | Placebo | | 100 mg<br>MIV-711 | | 200 mg<br>MIV-711 |
| | | Observed | Change | Observed | Change | Observed | Change |
| Visit | Statistic | N = x | N = x | N = x | N = x | N = x | N = x |
| | n | nn | | nn | | nn | |
| | Mean | xx.x | | xx.x | | XX.X | |
| VISIT 2 | SD | XX.XX | | xx.xx | | xx.xx | |
| Baseline | Median | XX.X | | XX.X | | XX.X | |
| | Min | XX | | XX | | XX | |
| | Max | xx | | xx | | xx | |
| | n | nn | nn | nn | nn | nn | nn |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| VISIT 5 | SD | XX.XX | xx.xx | XX.XX | xx.xx | XX.XX | XX.XX |
| WEEK 8 | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min | XX | XX | XX | XX | XX | XX |
| | Max | xx | XX | XX | XX | XX | XX |
| | n | nn | nn | nn | nn | nn | nn |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| VISIT 6 | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| WEEK 14 | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min | XX | XX | XX | XX | XX | XX |
| | Max | XX | XX | XX | XX | XX | XX |
| Etc | | | | | | | |

Programming note: table will be expanded to include all WOMAC stiffness questions

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Page X of Y

Medivir

Protocol Number: MIV-711-201

Parameter = Stiffness after First Woke Up in Morning

| | | | | Treati | ment | | |
|---|---|---|---|---|---|---|---|
| | | Place | Placebo | | 100 mg<br>MIV-711 | | 200 mg<br>MIV-711 |
| | | Observed | Change | Observed | Change | Observed | Change |
| Visit | Statistic | N = x | N = x | N = x | N = x | N = x | _ |
| VISIL | n | nn = x | N - X | nn | N - X | nn | N = X |
| | Mean | XX.X | | XX.X | | XX.X | |
| VISIT 2 | SD | XX.XX | | XX.XX | | XX.XX | |
| Baseline | Median | XX.X | | XX.X | | XX.X | |
| | Min | XX | | XX | | XX | |
| | Max | xx | | xx | | XX | |
| | n | nn | nn | nn | nn | nn | nn |
| | Mean | xx.x | xx.x | XX.X | xx.x | XX.X | XX.X |
| VISIT 5 | SD | XX.XX | xx.xx | xx.xx | xx.xx | xx.xx | XX.XX |
| WEEK 8 | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min | XX | XX | XX | XX | XX | XX |
| | Max | XX | XX | XX | XX | xx | XX |
| | n | nn | nn | nn | nn | nn | nn |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| VISIT 6 | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| WEEK 14 | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min | XX | XX | XX | XX | XX | XX |
| | Max | XX | XX | XX | XX | XX | XX |
| Etc | | | | | | | |

Programming note: table will be expanded to include all WOMAC Difficulty questions

Medivir

Final 1.0 Protocol: MIV-711-201 22 June 2017

Medivir

Protocol Number: MIV-711-201

Table 14.2.7 Number and Percentage of Patients with a Positive OARSI-OMERACT Response mITT Population

Parameter = Completely Better

| | Treatment | | |
|----------|------------|-------------------|-------------------|
| | Placebo | 100 mg<br>MIV-711 | 200 mg<br>MIV-711 |
| Response | N = x | N = X | N = x |
| Yes | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| No | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |


Page X of Y

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Page X of Y

Medivir

Protocol Number: MIV-711-201

Parameter = Knee Problem

| | _ | | Treatment | |
|---|---|---|---|---|
| Visit | | Placebo | 100 mg<br>MIV-711 | 200 mg<br>MIV-711 |
| | Score | N = x | N = x | N = x |
| | Completely better | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Much better | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| /ISIT 5 WEEK 8 | Better | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| VISII J WEEK O | No change | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Worse | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Much worse | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Completely better | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Much better | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| ISIT 6 WEEK 14 | Better | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| ISII O WEEK 14 | No change | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Worse | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Much worse | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Completely better | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Much better | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| ISIT 8 WEEK 26 | Better | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| IDII O WEEK 20 | No change | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Worse | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Much worse | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |

Programming note: table will be expanded to include all Global improvement questions: Knee Problem, Knee Pain, Ability to use knee.

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Page X of Y

Medivir

Protocol Number: MIV-711-201

Parameter = Mobility

| | | | | Treatr | ment | | |
|---|---|---|---|---|---|---|---|
| | | Placebo | | | 100 mg<br>MIV-711 | | 200 mg<br>MIV-711 |
| | | Observed | Change | Observed | Change | Observed | Change |
| Visit | Statistic | N = x | N = x | N = x | N = x | N = x | N = x |
| | n | nn | | nn | | nn | |
| | Mean | XX.X | | XX.X | | XX.X | |
| VISIT 2, | SD | XX.XX | | XX.XX | | XX.XX | |
| Day 1 | Median | XX.X | | XX.X | | XX.X | |
| | Min | XX | | XX | | XX | |
| | Max | XX | | xx | | xx | |
| | n | nn | nn | nn | nn | nn | nn |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | xx.x |
| VISIT 8 | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| WEEK 26 | Median | XX.X | XX.X | XX.X | xx.x | XX.X | XX.X |
| | Min | XX | XX | XX | XX | XX | XX |
| | Max | XX | XX | XX | XX | XX | XX |

Programming note: table will be expanded to include all QOL variables:
Mobility, self-care, usual activity, pain or discomfort, and anxiety or depression, health rating score.

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Page X of Y

Medivir

Protocol Number: MIV-711-201

Table 14.2.10.1

E-Diary NRS Scores Observed and Change from Baseline Summary, AM Reponse  $$\operatorname{\mathtt{mITT}}$  Population

Parameter = How would you rate overall pain severity over last 12 Hours?

| | | | | Treat | ment | | |
|---|---|---|---|---|---|---|---|
| | | Place | Placebo | | 100 mg<br>MIV-711 | | mg<br>711 |
| | | Observed | Change | Observed | Change | Observed | Change |
| Visit | Statistic | N = x | N = x | N = x | N = x | N = x | N = x |
| | n | nn | | nn | | nn | |
| | Mean | XX.X | | XX.X | | XX.X | |
| VISIT 2 | SD | XX.XX | | XX.XX | | XX.XX | |
| Baseline | Median | XX.X | | XX.X | | XX.X | |
| | Min | XX | | XX | | XX | |
| | Max | XX | | XX | | xx | |
| | n | nn | nn | nn | nn | nn | nn |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| VISIT 6 | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| WEEK 14 | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min | XX | XX | XX | XX | XX | XX |
| | Max | XX | XX | XX | XX | XX | XX |
| | n | nn | nn | nn | nn | nn | nn |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| VISIT 8 | SD | XX.XX | XX.XX | XX.XX | XX.XX | xx.xx | XX.XX |
| WEEK 26 | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min | XX | XX | XX | XX | XX | XX |
| | Max | XX | XX | XX | XX | XX | XX |

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Page X of Y

Medivir

Protocol Number: MIV-711-201

Table 14.2.10.2

E-Diary NRS Scores Observed and Change from Baseline Summary, PM Reponse  $$\operatorname{\mathtt{mITT}}$  Population

Parameter = How would you rate overall pain severity over last 12 Hours?

| | | | | Treat | ment | | |
|---|---|---|---|---|---|---|---|
| | | Place | Placebo | | 100 mg<br>MIV-711 | | mg<br>711 |
| | | Observed | Change | Observed | Change | Observed | Change |
| Visit | Statistic | N = x | N = x | N = x | N = x | N = x | N = x |
| | n | nn | | nn | | nn | |
| | Mean | XX.X | | XX.X | | XX.X | |
| VISIT 2 | SD | XX.XX | | XX.XX | | XX.XX | |
| Baseline | Median | XX.X | | XX.X | | XX.X | |
| | Min | XX | | XX | | XX | |
| | Max | XX | | XX | | xx | |
| | n | nn | nn | nn | nn | nn | nn |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| VISIT 6 | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| WEEK 14 | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min | XX | XX | XX | XX | XX | XX |
| | Max | XX | XX | XX | XX | XX | XX |
| | n | nn | nn | nn | nn | nn | nn |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| VISIT 8 | SD | XX.XX | XX.XX | XX.XX | XX.XX | xx.xx | xx.xx |
| WEEK 26 | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min | XX | XX | XX | XX | XX | XX |
| | Max | XX | XX | XX | XX | XX | XX |

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Page X of Y

Medivir

Protocol Number: MIV-711-201

Table 14.2.10.3

E-Diary NRS Scores Observed and Change from Baseline Summary, Overall Response  $$\operatorname{\mathtt{mITT}}$$  Population

Parameter = How would you rate overall pain severity over last 12 Hours?

| | | | | Treati | ment | | |
|---|---|---|---|---|---|---|---|
| | | Place | Placebo | | 100 mg<br>MIV-711 | | 200 mg<br>MIV-711 |
| | | Observed | Change | Observed | Change | Observed | Change |
| Visit | Statistic | N = x | N = x | N = x | N = x | N = x | N = x |
| | n | nn | | nn | | nn | |
| | Mean | XX.X | | XX.X | | XX.X | |
| VISIT 2 | SD | XX.XX | | XX.XX | | XX.XX | |
| Baseline | Median | XX.X | | XX.X | | XX.X | |
| | Min | XX | | XX | | XX | |
| | Max | XX | | xx | | xx | |
| | n | nn | nn | nn | nn | nn | nn |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| VISIT 6 | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| WEEK 14 | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min | XX | XX | XX | XX | XX | XX |
| | Max | XX | XX | xx | XX | xx | XX |
| | n | nn | nn | nn | nn | nn | nn |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| VISIT 8 | SD | XX.XX | XX.XX | xx.xx | xx.xx | xx.xx | xx.xx |
| WEEK 26 | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min | XX | XX | XX | XX | XX | XX |
| | Max | XX | XX | XX | XX | XX | XX |

Programming note: The mean of the AM, PM NRS scores will be used to obtain 1 record at each visit prior to computing descriptive statistics

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Page X of Y

Medivir

Protocol Number: MIV-711-201

Table 14.2.10.4

Number and Percentage of Patients with E-Diary Pain Medication Usage (Yes/No) Over Last 12 Hours, AM Response

mITT Population

Question = Have you taken any pain medication over the last 12 hours since you last answered your OA Daily Diary?

| | | | Treatment | |
|---|---|---|---|---|
| Visit | | Placebo | 100 mg<br>MIV-711 | 200 mg<br>MIV-711 |
| | Score | N = x | N = x | N = x |
| VISIT 2 Baseline | Yes | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| VISII 2 Daseiine | No | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| VISIT 6 WEEK 14 | Yes | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| VIDII O WEEK 14 | No | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| VISIT 8 WEEK 26 | Yes | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| VISII O WEEK 20 | No | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Page X of Y

Medivir

Protocol Number: MIV-711-201

Table 14.2.10.5

Number and Percentage of Patients with E-Diary Pain Medication Usage (Yes/No) Over Last 12 Hours, PM Response mITT Population

Question = Have you taken any pain medication over the last 12 hours since you last answered your OA Daily Diary?

| | | Treatment | | |
|---|---|---|---|---|
| Visit | | Placebo | 100 mg<br>MIV-711 | 200 mg<br>MIV-711 |
| | Score | N = x | N = x | N = x |
| VISIT 2 Baseline | Yes | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| VIDII Z BASCIINC | No | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| VISIT 6 WEEK 14 | Yes | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| VIDII O WEEK 14 | No | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| VISIT 8 WEEK 26 | Yes | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| VISII O WEEK 20 | No | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |

Medivir

Protocol: MIV-711-201 22 June 2017

Medivir Page X of Y

Protocol Number: MIV-711-201

Table 14.2.10.6

Number and Percentage of Patients with E-Diary Pain Medication Usage (Yes/No) Over Last 12 Hours, Overall Response mITT Population

Question = Have you taken any pain medication over the last 12 hours since you last answered your OA Daily Diary?

| | | | Treatment | |
|---|---|---|---|---|
| Visit | | Placebo | 100 mg<br>MIV-711 | 200 mg<br>MIV-711 |
| | Score | N = x | N = x | N = x |
| VISIT 2 Baseline | Yes | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| VIDIT 2 DASCIINC | No | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| VISIT 6 WEEK 14 | Yes | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| VIOIT O WHEN IT | No | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| VISIT 8 WEEK 26 | Yes | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| VISII O WEEK 20 | No | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |

Programming note: at least one 'Yes' response for AM or PM will be interpreted as a 'Yes' response 24 hours overall.

Final 1.0

Medivir Protocol: MIV-711-201 Final 1.0 22 June 2017

Table 14.2.10.7
E-Diary Pain Medication Usage Over Last 12 Hours
Number and Percentage of Patients with each Reported Category, AM Response mITT Population

| | - | Treatment | | |
|---|---|---|---|---|
| Visit | | Placebo | 100 mg<br>MIV-711 | 200 mg<br>MIV-711 |
| | Category | N = x | N = x | N = x |
| | Less than Normal | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| VISIT 2, Baseline | Normal | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | More than Normal | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Less than Normal | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| VISIT 6 WEEK 14 | Normal | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | More than Normal | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Less than Normal | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| VISIT 8 WEEK 26 | Normal | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | More than Normal | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |

Medivir

Protocol: MIV-711-201 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Final 1.0

# Table 14.2.10.8 E-Diary Pain Medication Usage Over Last 12 Hours Number and Percentage of Patients with each Reported Category, PM Response mITT Population

| | | | Treatment | |
|---|---|---|---|---|
| Visit | | Placebo | 100 mg<br>MIV-711 | 200 mg<br>MIV-711 |
| | Category | N = x | N = x | N = x |
| | Less than Normal | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| VISIT 2, Baseline | Normal | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | More than Normal | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Less than Normal | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| VISIT 6 WEEK 14 | Normal | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | More than Normal | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Less than Normal | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| VISIT 8 WEEK 26 | Normal | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | More than Normal | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |

Medivir

Final 1.0 Protocol: MIV-711-201 22 June 2017

Medivir

Page X of Y Protocol Number: MIV-711-201

Table 14.3.1.1 Summary of Treatment Emergent Adverse Events SAF Population

| | | Treatment | | - |
|---|---|---|---|---|
| | Placebo<br>N = x<br>nn (%) E | 100 mg<br>MIV-711<br>N = x<br>nn (%) E | 200 mg<br>MIV-711<br>N = x<br>nn (%) E | Overall N = x nn (%) E |
| All AEs | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E |
| 'Related' AEs | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E |
| Mild AEs | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E |
| Moderate AEs | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E |
| Severe AEs | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E |
| Deaths | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E |
| Serious AEs | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E |
| AEs Leading to early discontinuation from study | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E |

TEAE = Treatment Emergent Adverse Event nn = Number of Patientswith TEAEs

N = Number of PatientsExposed

 $(nn.n%) = nn/N \times 100$ E = Number of AEs

Medivir
Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Table 14.3.1.2

Number and Percentage of Patients with Treatment Emergent Adverse Events by System Organ Class, Preferred Term, and Treatment SAF Population

| | | Treatment | | _ |
|---|---|---|---|---|
| System Organ Class Preferred Term | Placebo | 100 mg<br>MIV-711 | 200 mg<br>MIV-711 | Overall |
| | N = x | N = x | N = x | N = x |
| System Organ Class 1 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term 1 | , , | , , | , , , , , | , , |
| | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term 2 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term 3 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term xx | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| System Organ Class 2 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term 1 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term 2 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term 3 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term xx | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |

Medivir

Final 1.0 Protocol: MIV-711-201 22 June 2017

Medivir

Protocol Number: MIV-711-201

Table 14.3.1.3

Number and Percentage of Patients with Treatment Emergent Adverse Events 'Related to IMP' by System Organ Class, Preferred Term, Severity, and Treatment SAF Population

| | | | Treatment | | |
|---|---|---|---|---|---|
| System Organ Class Preferred Term | Severity | Placebo | 100 mg<br>MIV-711 | 200 mg<br>MIV-711 | Overall N = x |
| lielelled leim | Severicy | N = x | N = x | N = x | IV — X |
| System Organ Class 1 | Mild | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Moderate | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Severe | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term 1 | Mild | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Moderate | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Severe | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term xx | Mild | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Moderate | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Severe | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| System Organ Class 2 | Mild | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Moderate | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Severe | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term 1 | Mild | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Moderate | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Severe | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term xx | Mild | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Moderate | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Severe | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Etc | | | | | |

For patients with multiple adverse events of the same preferred term and different severities, the AE with the highest assessment of severity was used in the summary table.

Page X of Y

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Page X of Y

Medivir

Protocol Number: MIV-711-201

Table 14.3.1.4

Number and Percentage of Patients with Treatment Emergent Adverse Events 'Not Related to IMP' by System Organ Class, Preferred Term, Severity, and Treatment

SAF Population

| | | | Treatment | | |
|---|---|---|---|---|---|
| | | Placebo | 100 mg | 200 mg | Overall |
| System Organ Class | | | MIV-711 | MIV-711 | |
| Preferred Term | Severity | | | | N = X |
| | | N = X | N = x | N = x | |
| System Organ Class 1 | Mild | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Moderate | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Severe | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term 1 | Mild | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Moderate | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Severe | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term xx | Mild | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Moderate | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Severe | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| System Organ Class 2 | Mild | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Moderate | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Severe | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term 1 | Mild | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Moderate | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Severe | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term xx | Mild | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Moderate | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Severe | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Etc | | | | | |

For patients with multiple adverse events of the same preferred term and different severities, the AE with the highest assessment of severity was used in the summary table.

Medivir
Protocol: MIV-711-201
22 June 2017

Medivir Page X of Y

Protocol Number: MIV-711-201

Table 14.3.1.5

Number and Percentage of Patients with Serious Treatment Emergent Adverse Events by System Organ Class, Preferred Term, and Treatment SAF Population

| | | Treatment | | |
|---|---|---|---|---|
| System Organ Class Preferred Term | Placebo | 100 mg<br>MIV-711 | 200 mg<br>MIV-711 | Overall |
| | N = x | N = x | N = x | N = x |
| System Organ Class 1 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term 1 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term 2 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term 3 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term xx | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| System Organ Class 2 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term 1 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term 2 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term 3 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term xx | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |

Medivir

Final 1.0 Protocol: MIV-711-201 22 June 2017

Medivir

Protocol Number: MIV-711-201

Table 14.3.1.6

Number and Percentage of Patients with Treatment Emergent Adverse Events Leading to Discontinuation by System Organ Class, Preferred Term, and Treatment SAF Population

| | | Treatment | | |
|---|---|---|---|---|
| System Organ Class Preferred Term | Placebo | 100 mg<br>MIV-711 | 200 mg<br>MIV-711 | Overall |
| riciciica icim | N = x | N = x | N = x | N = x |
| System Organ Class 1 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term 1 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term 2 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term 3 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term xx | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| System Organ Class 2 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term 1 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term 2 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term 3 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term xx | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |

Page X of Y

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Page X of Y

Medivir

Protocol Number: MIV-711-201

Table 14.3.2.1

Clinical Laboratory Chemistry - Summary of Observed Values
SAF Population

Lab Parameter = Lab Parameter (unit)

| | | | Treatment | | - |
|---|---|---|---|---|---|
| | | Placebo | 100 mg<br>MIV-711 | 200 mg<br>MIV-711 | Overall |
| Visit | Statistic | N = x | N = x | N = x | N = x |
| | n | nn | nn | nn | nn |
| | Mean | XX.X | XX.X | XX.X | XX.X |
| Screening | SD | xx.xx | xx.xx | xx.xx | XX.XX |
| | Median | xx.x | xx.x | xx.x | XX.X |
| | Min | XX | xx | xx | XX |
| | Max | XX | XX | XX | XX |
| | n | nn | nn | nn | nn |
| Visit 2 | Mean | XX.X | xx.x | xx.x | XX.X |
| Baseline | SD | XX.XX | xx.xx | xx.xx | XX.XX |
| Day 1 | Median | XX.X | XX.X | XX.X | XX.X |
| Jay I | Min | XX | xx | xx | XX |
| | Max | XX | XX | XX | XX |
| | n | nn | nn | nn | nn |
| | Mean | XX.X | XX.X | XX.X | XX.X |
| /isit 3 | SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Week 2 | Median | XX.X | XX.X | XX.X | XX.X |
| | Min | XX | XX | XX | XX |
| | Max | XX | XX | XX | XX |
| | n | nn | nn | nn | nn |
| Visit 4 | Mean | XX.X | XX.X | XX.X | XX.X |
| Veek 4 | SD | XX.XX | xx.xx | xx.xx | XX.XX |
| VCCA 1 | Median | XX.X | xx.x | XX.X | XX.X |
| | Min | XX | xx | xx | XX |
| | Max | XX | xx | xx | XX |
| Etc | | | | | |

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Page X of Y

Medivir

Protocol Number: MIV-711-201

Table 14.3.2.2 Clinical Laboratory Hematology - Summary of Observed Values SAF Population

Lab Parameter = Lab Parameter (unit)

| | | | Treatment | | |
|---|---|---|---|---|---|
| | | Placebo | 100 mg<br>MIV-711 | 200 mg<br>MIV-711 | Overall |
| Visit | Statistic | N = x | N = x | N = x | N = x |
| | n | nn | nn | nn | nn |
| | Mean | XX.X | xx.x | xx.x | XX.X |
| Screening | SD | xx.xx | xx.xx | xx.xx | XX.XX |
| | Median | XX.X | xx.x | xx.x | XX.X |
| | Min | XX | xx | xx | XX |
| | Max | XX | XX | XX | XX |
| | n | nn | nn | nn | nn |
| Jisit 2 | Mean | XX.X | xx.x | xx.x | XX.X |
| Baseline | SD | XX.XX | xx.xx | xx.xx | XX.XX |
| Day 1 | Median | XX.X | xx.x | XX.X | XX.X |
| Jay I | Min | XX | XX | XX | XX |
| | Max | XX | XX | XX | XX |
| | n | nn | nn | nn | nn |
| | Mean | XX.X | XX.X | XX.X | XX.X |
| 7isit 3 | SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Week 2 | Median | XX.X | XX.X | XX.X | XX.X |
| | Min | XX | XX | XX | XX |
| | Max | XX | XX | XX | XX |
| | n | nn | nn | nn | nn |
| Jisit 4 | Mean | XX.X | XX.X | XX.X | XX.X |
| Veek 4 | SD | XX.XX | xx.xx | xx.xx | XX.XX |
| .ccx i | Median | XX.X | xx.x | xx.x | XX.X |
| | Min | XX | xx | xx | XX |
| | Max | XX | XX | XX | XX |
| Etc | | | | | |

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Page X of Y

Medivir

Protocol Number: MIV-711-201

Table 14.3.2.3

Clinical Laboratory Chemistry - Shift From Baseline to Maximum Post-dose Value SAF Population

Lab Parameter = Lab Parameter (unit)

| | | Baseline (Visit 2) | | | | | |
|---|---|---|---|---|---|---|---|
| | Maximum | | Low | N | Normal | | High |
| Treatment | Post-dose | | | | | | |
| | Value | | | | | | |
| | Low | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| Placebo | Normal | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| | High | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| | Low | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| 100 mg | Normal | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| MIV-711 | High | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| | Low | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| 200 mg | Normal | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| MIV-711 | High | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| | = | | | | | | |

Programming Note: Similar table will be created for hematology parameters: Tables 14.3.2.4

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Page X of Y

Medivir

Protocol Number: MIV-711-201

Table 14.3.2.5

Clinical Laboratory Chemistry - Shift From Baseline to Minimum Post-dose Value SAF Population

Lab Parameter = Lab Parameter (unit)

| | | Baseline (Visit 2) | | | | | |
|---|---|---|---|---|---|---|---|
| | Maximum | | Low | 1 | Normal | | High |
| Treatment | Post-dose | | | | | | |
| | Value | | | | | | |
| | Low | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| Placebo | Normal | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| | High | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| | Low | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| 100 mg | Normal | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| MIV-711 | High | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| | Low | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| 200 mg | Normal | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| MIV-711 | High | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| | 2 | | | | | | . , |

Programming Note: Similar table will be created for hematology parameters: Tables 14.3.2.6

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Page X of Y

Medivir

Protocol Number: MIV-711-201

Table 14.3.3

 $\hbox{ Vital Signs Blood Pressure and Heart Rate Summary of Observed and Change from Baseline Values } \\ \hbox{ SAF Population}$ 

Parameter = Systolic Blood Pressure (mmHg)

| | | | | Treatr | nent | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | 100 mg | | 200 | mg | Overa | a⊥⊥ |
| | | Place | ebo | MIV- | 711 | MIV- | 711 | Ν - | |
| | | | | | | | | N = x | |
| | | Observed | Change | Observed | Change | Observed | Change | Observed | Chang |
| Visit | Statistic | N = x | N = x | N = x | N = x | N = x | N = x | N = x | N = > |
| | n | nn | nn | nn | nn | nn | nn | nn | nn |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Screening | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Median | XX.X | XX.X | XX.X | xx.x | XX.X | XX.X | XX.X | XX.X |
| | Min | XX | XX | XX | XX | XX | XX | XX | XX |
| | Max | XX | XX | XX | XX | XX | XX | XX | XX |
| | n | nn | nn | nn | nn | nn | nn | nn | nn |
| Visit 2 | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Baseline | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.X |
| Day 1 | Median | XX.X | XX.X | XX.X | xx.x | XX.X | XX.X | XX.X | XX.X |
| | Min | XX | XX | XX | XX | XX | XX | XX | XX |
| | Max | XX | XX | XX | XX | XX | XX | XX | XX |
| | n | nn | nn | nn | nn | nn | nn | nn | nn |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX. |
| Visit 3 | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.X |
| Week 2 | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min | XX | XX | XX | XX | XX | XX | XX | XX |
| | Max | XX | XX | XX | XX | XX | XX | XX | XX |

Programming Notes: Table will be expanded to include diastolic blood pressure and heart rate, subject weight

Medivir

Protocol: MIV-711-201 22 June 2017

Medivir

Protocol Number: MIV-711-201

Table 14.3.4.1

12 Lead ECG - Summary of Observed and Change from Baseline Values

SAF Population

Parameter = QT Interval (unit)

| | | Treatment | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | 100 mg 200 mg Placebo MIV-711 MIV-711 | | Over | all | | | | |
| | | Placebo | | rii v | MIT A — \ T T | | MI V - 7 I I | | N = x |
| | | Observed | Change | Observed | Change | Observed | Change | Observed | Change |
| Visit | Statistic | N = x | N = x | N = x | N = x | N = x | N = x | N = x | N = x |
| | n | nn | nn | nn | nn | nn | nn | nn | nn |
| | Mean | XX.X | xx.x | XX.X | xx.x | XX.X | xx.x | XX.X | xx.x |
| Screening | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | xx.x |
| | Min | XX | XX | XX | XX | XX | XX | XX | XX |
| | Max | XX | XX | xx | XX | XX | XX | xx | XX |
| | n | nn | nn | nn | nn | nn | nn | nn | nn |
| Visit 2 | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Baseline | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Day 1 | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | xx.x |
| | Min | XX | XX | XX | XX | XX | XX | XX | XX |
| | Max | XX | XX | XX | XX | XX | XX | XX | XX |
| | n | nn | nn | nn | nn | nn | nn | nn | nn |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Visit 3 | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Week 2 | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min | XX | XX | XX | XX | XX | XX | XX | XX |
| | Max | XX | XX | XX | XX | XX | XX | XX | XX |
| Etc | | | | | | | | | |

QTcB = QT corrected according to Bazett, QTcF = QT corrected according to Fridericia.

Programming note: Table will include: QTcB interval and QTcF interval

Final 1.0

Page X of Y

Medivir

Final 1.0 Protocol: MIV-711-201 22 June 2017

Medivir

Protocol Number: MIV-711-201

Table 14.3.4.2 12 Lead ECG - Categorical Summary of Observed Values

> SAF Population Parameter = QT (msec)

| | | | Treatment | | - |
|---|---|---|---|---|---|
| Visit | | Placebo | 100 mg<br>MIV-711 | 200 mg<br>MIV-711 | Overall |
| | Category (unit) | | | | N = X |
| | | N = x | N = x | N = x | |
| | ≤ 450 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Screening | $450 < to \le 480$ | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Screening | $480 < to \le 500$ | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | >500 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | ≤ 450 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Visit 2 Baseline Day 1 | $450 < to \le 480$ | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| visic 2 baseline bay i | $480 < to \le 500$ | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | >500 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | ≤ 450 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Visit 3 Week 2 | $450 < to \le 480$ | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| visic 3 week 2 | $480 < to \le 500$ | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | >500 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Etc | Etc | | | | |

 ${\tt QTcB} = {\tt QT}$  corrected according to Bazett,  ${\tt QTcF} = {\tt QT}$  corrected according to Fridericia.

Programming note: Table will include: QTcB interval and QTcF interval

Page X of Y

Medivir

Final 1.0 Protocol: MIV-711-201 22 June 2017

Medivir Page X of Y

Protocol Number: MIV-711-201

#### Table 14.3.4.3 12 Lead ECG - Categorical Summary of Change from Baseline SAF Population

Parameter = QT (msec)

| | | | Treatment | | _ |
|---|---|---|---|---|---|
| Visit | Category (unit) | Placebo | 100 mg<br>MIV-711 | 200 mg<br>MIV-711 | Overall |
| | | N = x | N = x | N = x | N = x |
| | <= 0 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Visit 3 Week 2 | >0 to ≤ 30 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| VISIC 5 WCCK 2 | >30 to ≤ 60 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | >60 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | <= 0 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Visit 4 Week 4 | >0 to ≤ 30 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | >30 to ≤ 60 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | >60 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Etc | | | | | |

QTcB = QT corrected according to Bazett, QTcF = QT corrected according to Fridericia.

Programming note: Table will include: QTcB interval and QTcF interval

Medivir
Protocol: MIV-711-201
22 June 2017

15. Listing Shells

Medivir
Protocol: MIV-711-201
22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Listing 16.2.1.1 Patient Disposition

| Patient | Completion Status | If Discontinued,<br>Day of<br>Withdrawal | If Discontinued,<br>Date of<br>Withdrawal | Reason For<br>Discontinuation | Finalization<br>of Visit 9<br>(Week 30) | Roll-over to<br>and<br>finalization<br>of Visit 2 of<br>MIV-711-202 |
|---|---|---|---|---|---|---|
| | Completed<br>Discontinued | | | | | |

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Listing 16.2.1.2 Patients Excluded from the Analysis Populations

| Patient | Population | Reason for Exclusion |
|---------|------------|----------------------|
| | ITT | |
| | mITT | |
| | PPS | |
| | SAF | |

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Listing 16.2.1.3 Enrolled Patients Who Did Not Meet All Eligibility Criteria

| Patient | Criteria Category | Criteria Description | Response |
|---------|-------------------|----------------------|----------|
| | Inclusion | | No |
| | Exclusion | | Yes |

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Listing 16.2.1.4
Exclusion Tests
FSH test, Serology, Urine Drug Screen

Treatment = MIV-711 200 mg

Collection Collection

Patient Visit Date Time Exclusion Test Result Units

FSH test

Etc...

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Listing 16.2.2.1 Protocol Deviations

| | Study | | Date Deviation | ~ . | | |
|---|---|---|---|---|---|---|
| Patient | Day | Time Point | Occurred | Category | Explanation | Classification |
| | | | | Time Windo | w | Minor |
| | | | | Dosing | | Major |
| | | | | Exclusion Te | ests | Major |
| | | | | Etc | | |
Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Listing 16.2.4.1 Demographics

Treatment = MIV-711 200 mg

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Listing 16.2.4.2 Medical History

Treatment = MIV-711 200 mg

Reported Term >MedDRA Preferred

Term

>>System Organ
Patient Class

Onset Date

Status

Recovered Date Currently Treated with Medication?

Ongoing Yes/No

Medivir

Final 1.0 Protocol: MIV-711-201 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Listing 16.2.5.1 Prior and Concomitant Medications

Treatment = MIV-711 200 mg

Medication Name Was >WHO Drug Name Pain Start Dose/ There Stop >>ATC Medication Unit Frequency Route Indication an AE Patient Classification Category Date Date Ongoing? Prior Yes/No Yes/No CM

Programming note: Pain Medication = 'Yes' if ATC = 'ANALGESICS'

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Listing 16.2.5.2
Dose Administration

Treatment = MIV-711 200 mg

Date of Time of Dose Form / Category of Patient Visit Dose Dose Route Treatment

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Listing 16.2.5.3
Dose Administration Compliance

Treatment = MIV-711 200 mg

| | | | | | | | | | | Reason | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | Actual | | Were all | not all | | Number | |
| | | | | | | | Number | Planned | unused | unused | | of Days | |
| | | Date | Time | Category | Dispensed | Returned | of | number | Capsules | Capsules | Medication | exposed | IMP |
| | | of | of | of | Amount | Amount | Capsules | of | returned? | returned | error | to IMP | Compliance |
| Patient | Visit | Dose | Dose | Treatment | (Capsules) | (Capsules) | used | capsules | | | | | _ |

The 'actual number of capsules used' was derived as the 'number of capsules dispensed' minus the 'number of capsules returned'.

'Planned number of capsules' is the number of days of per protocol dosing from V2 (first dose) to V8 (last dose), since each patient is to receive 1 capsule of dosing per day of dose administration.

IMP compliance: (actual number of capsules used / planned number of capsules administered)  $\times$  100%

Medivir

Final 1.0 Protocol: MIV-711-201 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Listing 16.2.6.1 Numerical Rating Scale of Knee Pain

Treatment = MIV-711 200 mg

| | | | | Pain | | | | |
|---|---|---|---|---|---|---|---|---|
| | | | | Severity | | | | |
| | | | Target | in | | Satisfied | Worst | Overall |
| | | | Knee | Target | | with | Pain | pain |
| | | | Used | Knee | Global | Target | Severity | severity |
| | | Date of | for | (last | Assessment | Knee | Target | in other |
| Patient | Visit | Assessment | NRS | week) | NRS | Function | Knee | knee |

VISIT 2 BASELINE DAY VISIT 5 WEEK 8 VISIT 6 WEEK 14 Etc...

Programming note: listing will include:

- Primary endpoint: Amount of pain severity in the target knee last week (SDTM: Overall pain severity in target knee
- Global Assessment Score: How active has the target knee arthritis has been in the past week (SDTM: How active was target knee arthritis)
- Satisfaction with target knee function (SDTM: How satisfied are you with target knee function)
- Worst pain severity in target knee (SDTM: Worst pain severity in target knee)
- Overall pain severity in other knee (SDTM: Overall pain severity in other knee)

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

#### Listing 16.2.6.2 Numerical Rating Scale of Knee Pain Change From Baseline

Treatment = MIV-711 200 mg

| • | | | Pain | | | | |
|---|---|---|---|---|---|---|---|
| | | | Severity | | | | |
| | | | in | | Satisfied | Worst | Overall |
| | | | Target | | with | Pain | pain |
| | | | Knee | Global | Target | Severity | severity |
| | | Date of | (last | Assessment | Knee | Target | in other |
| Patient | Visit | Assessment | week) | NRS | Function | Knee | knee |

VISIT 2 BASELINE DAY VISIT 5 WEEK 8 VISIT 6 WEEK 14 Etc...

Programming note: listing will include:

- Primary endpoint: Amount of pain severity in the target knee last week (SDTM: Overall pain severity in target knee
- Global Assessment Score: How active has the target knee arthritis has been in the past week (SDTM: How active was target knee arthritis)
- Satisfaction with target knee function (SDTM: How satisfied are you with target knee function)
- Worst pain severity in target knee (SDTM: Worst pain severity in target knee)
- Overall pain severity in other knee (SDTM: Overall pain severity in other knee)

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Treatment = MIV-711 200 mg

Duration
of
Knee
Pain
Past
Date of 12 Onset of
Patient Visit Assessment Months Knee Pain

VISIT 2 BASELINE DAY VISIT 5 WEEK 8

VISIT 6 WEEK 14

Etc...

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Listing 16.2.6.4

Imaging Results - MRI of Bone Area for the Target Knee
Observed and Change from Baseline

Treatment = MIV-711 200 mg

MRI MRI Result Result Change from
Date of Time of - Bone baseline
Patient Visit Assessment Assessment area Bone Area

VISIT 2 BASELINE DAY VISIT 8 WEEK 26

Programming note: source data obtained from MF\_TAB: Area of bone in the medial femur region, MF

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Listing 16.2.6.5

Imaging Results - MRI of Cartilage Thickness for the Target Knee
Observed and Change from Baseline

Treatment = MIV-711 200 mg

MRI Result
- Change
MRI from
MRI from
ResultDate of Time of Cartilage
Patient Visit Assessment Region Thickness Thickness

VISIT 2 BASELINE DAY VISIT 8 WEEK 26

Programming note: source data obtained from:

- CM FEMUR THCTAB: Average thickness of cartilage in the central medial femur region
- CM TIBIA THCTAB: Average thickness of cartilage in the central medial tibia region

Medivir

Protocol: MIV-711-201

Medivir

Page X of Y Protocol Number: MIV-711-201

Etc...

Listing 16.2.6.6
Other Secondary Imaging Variables - MOAKS

Treatment = MIV-711 200 mg

| Patient | Visit | Date of<br>Assessment | Time of<br>Assessment | Question<br>Group Name | Question<br>Sub-Group<br>Name | Question Name | Result<br>Score | Result<br>Score<br>Description | Comments |
|---|---|---|---|---|---|---|---|---|---|
| | VISIT 2 BASELINE DAY VISIT 8 WEEK 26 | | | BML and<br>Cyst | Size of<br>BML | Medial Patella | | | |
| | | | | | | Lateral Patella<br>Medical Femur<br>Trochlea<br>Etc | | | |
| | | | | | Number of<br>BMLs | Medial Patella | | | |
| | | | | | | Lateral Patella<br>Medical Femur<br>Trochlea<br>Etc | | | |
| | | | | | Percent<br>that is<br>BML | Medial Patella | | | |
| | | | | | | Lateral Patella<br>Medical Femur<br>Trochlea<br>Etc | | | |
| | | | | Cartilage<br>Assessment | | Medial Patella | | | |
| | | | | | | Lateral Patella<br>Medical Femur<br>Trochlea | | | |

Etc..

Etc...

Final 1.0 22 June 2017

Medivir

Protocol: MIV-711-201 22 June 2017

Medivir Page X of Y

Protocol Number: MIV-711-201 Listing 16.2.6.7

Other Secondary Imaging Variables Change from Baseline - MOAKS

Treatment = MIV-711 200 mg

| Patient | Visit | Date of<br>Assessment | Time of<br>Assessment | Question<br>Group Name | Question<br>Sub-Group<br>Name | Question Name | Change<br>Score |
|---|---|---|---|---|---|---|---|
| | VISIT 2 BASELINE DAY<br>VISIT 8 WEEK 26 | | | BML and<br>Cyst | Size of<br>BML | Medial Patella | |
| | | | | | | Lateral Patella | |
| | | | | | | Medical Femur<br>Trochlea<br>Etc | |
| | | | | | Number of<br>BMLs | Medial Patella | |
| | | | | | | Lateral Patella<br>Medical Femur<br>Trochlea<br>Etc | |
| | | | | | Percent<br>that is<br>BML | Medial Patella | |
| | | | | | | Lateral Patella<br>Medical Femur<br>Trochlea<br>Etc | |
| | | | | Cartilage<br>Assessment | Size of<br>Cartilage<br>Loss | Medial Patella | |
| | | | | | | Lateral Patella<br>Medical Femur<br>Trochlea | |
| | | | | Etc | Etc | Etc | |

Programming note: only select variables will be considered for change from baseline calculation per sponsor request. Will be noted in final SAP text.

Final 1.0

Medivir

Protocol: MIV-711-201

Page X of Y

Final 1.0

22 June 2017

Medivir

Protocol Number: MIV-711-201

Listing 16.2.6.8

Other Secondary Imaging Variables - Imorphics

Treatment = MIV-711 200 mg

| Patient | Visit | Date of<br>Assessment | Time of<br>Assessment | Question<br>Group Name | ~ | Question Name | Result<br>Score | Result<br>Score<br>Description | Comments |
|---|---|---|---|---|---|---|---|---|---|
| V | ISIT 2 | | | | | | | | |

BASELINE DAY VISIT 8 WEEK 26

Medivir

Protocol: MIV-711-201

Page X of Y Medivir

Protocol Number: MIV-711-201

Listing 16.2.6.9
Other Secondary Imaging Variables Change from Baseline - Imorphics

Treatment = MIV-711 200 mg

| Patient | Visit | Date of<br>Assessment | Time of<br>Assessment | Question<br>Group Name | Question<br>Sub-Group<br>Name | Question Name | Change<br>Score |
|---|---|---|---|---|---|---|---|
| | VISIT 2 | | | | | | |

BASELINE DAY VISIT 8 WEEK 26

Final 1.0

22 June 2017

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Listing 16.2.6.10
Observed Raw ICOAP Scores

Treatment = MIV-711 200 mg

Date of Time of
Patient Visit Assessment Assessment IP1 IP2 IP3 IP4 IP5 IP6 IP9 IP9 IP9

VISIT 2 BASELINE DAY

VISIT 5 WEEK 8 VISIT 6 WEEK 14

Etc...

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Listing 16.2.6.11
Transformed ICOAP Scores

Treatment = MIV-711 200 mg

Intermittent pain

Constant Pain Subscale subscale

Total pain score

Date of Time of
Patient Visit Assessment Assessment Observed Change Observed Change
VISIT 2 BASELINE
DAY

VISIT 5 WEEK 8 VISIT 6 WEEK 14

Etc...

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

| | | | Walking | Going | | Sitting | |
|---|---|---|---|---|---|---|---|
| | | Date | on | Up or | at Night | or | |
| | | Of | a Flat | Down | While | Lying | While |
| Patient | Visit | Assessment | Surface | Stairs | in Bed | Down | Standing |

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Listing 16.2.6.13
Western Ontario and McMaster Index (WOMAC) - Stiffness Questions

| | | | Stiffness | |
|---------|-------|------------|-----------|-----------|
| | | | after | |
| | | | First | Stiffness |
| | | Date | Woke Up | Sitting |
| | | Of | in | or Lying |
| Patient | Visit | Assessment | Morning | Down |

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Treatment = MIV-711 200 mg

| | | | When | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | | going | When | Getting | | When | Walking |
| | | Date | Down | Going | Up | | Bending | on |
| | | Of | the | Up the | from a | While | to the | a Flat |
| Patient | Visit | Assessment | Stairs | Stairs | sitting | Standing | Floor | Surface |

Programming note: listing will be expanded to show all 17 difficulty questions

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Listing 16.2.6.15

Western Ontario and McMaster Index (WOMAC) Change from Baseline - Pain Questions

| | | | Walking | Going | | Sitting | |
|---|---|---|---|---|---|---|---|
| | | Date | on | Up or | at Night | or | |
| | | Of | a Flat | Down | While | Lying | While |
| Patient | Visit | Assessment | Surface | Stairs | in Bed | Down | Standing |

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

| | | | Stiffness | |
|---------|-------|------------|-----------|-----------|
| | | | after | |
| | | | First | Stiffness |
| | | Date | Woke Up | Sitting |
| | | Of | in | or Lying |
| Patient | Visit | Assessment | Morning | Down |

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Listing 16.2.6.17

Western Ontario and McMaster Index (WOMAC) Change from Baseline - Difficulty Questions

Treatment = MIV-711 200 mg

| | | | When | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | | going | When | Getting | | When | Walking |
| | | Date | Down | Going | Up | | Bending | on |
| | | Of | the | Up the | from a | While | to the | a Flat |
| Patient | Visit | Assessment | Stairs | Stairs | sitting | Standing | Floor | Surface |

Programming note: listing will be expanded to show all 17 difficulty questions

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Listing 16.2.6.18

OARSI-OMERACT Responder Index
Derived Scores out of 100

Treatment = MIV-711 200 mg

| Total Total WOMAC WOMAC Pain Function WOMAC Pair Score Score Score Patient Visit [1] [2] 100 | Global Global Assessment Score NRS 100 100 |
|---|---|
|---|---|

Visit 2 Visit 8

- [1] Total WOMAC Pain Score (Total\_WOMAC\_Pain\_50): sum of the 5 WOMAC pain responses
  [2] Total WOMAC Function Score (Total\_WOMAC\_Func\_170): sum of the 17 WOMAC function responses
  Global Assessment NRS = "How Active Target Knee Arthritis Has Been", from Listing 16.2.6.1
- WOMAC PAIN Score 100 = Total\_WOMAC\_Pain\_50 x 2. WOMAC Function Score 100 = Total\_WOMAC\_Func\_170  $\div$  1.7. Global Assessment NRS 100= (Global Assessment NRS) x 10.

Medivir

Protocol: MIV-711-201 22 June 2017

Medivir
Protocol Number: MIV-711-201
Page X of Y

Listing 16.2.6.19

OARSI-OMERACT Responder Index

Change from Baseline and Percentage Change from Baseline Scores

Treatment = MIV-711 200 mg

| | | Change<br>From | Percent<br>Change From | | Response | |
|---|---|---|---|---|---|---|
| Patient | Score | Baseline | Baseline | Criteria | per Score | Responder |
| 101 | WOMAC Pain Score 100 | XX | уу | | No | No |
| 101 | WOMAC Function Score 100 | XX | УУ | | No | |
| 101 | Global Assessment NRS 100 | XX | УУ | 5 | No | |
| 102 | WOMAC Pain Score 100 | XX | УУ | 1 | Yes | Yes |
| 102 | WOMAC Function Score 100 | XX | УУ | 2 | Yes | |
| 102 | Global Assessment NRS 100 | XX | УУ | | No | |
| 103 | WOMAC Pain Score 100 | XX | УУ | 3 | Yes | Yes |
| 103 | WOMAC Function Score 100 | XX | УУ | | No | |
| 103 | Global Assessment NRS 100 | XX | УУ | 5 | Yes | |
| 104 | WOMAC Pain Score 100 | XX | УУ | 3 | Yes | |
| 104 | WOMAC Function Score 100 | XX | УУ | 4 | Yes | |
| 104 | Global Assessment NRS 100 | XX | УУ | | No | |
| 105 | WOMAC Pain Score 100 | XX | УУ | | No | |
| 105 | WOMAC Function Score 100 | XX | УУ | 4 | No | |
| 105 | Global Assessment NRS 100 | XX | УУ | | No | |

Percent Change from Baseline: ((Visit 8 Score - Visit 2 Score) ÷ Visit 2 Score) x 100

Criteria 1: WOMAC Pain: decrease from baseline >=20 and Percentage Decrease from Baseline >=50%

Criteria 2: WOMAC Function: decrease from baseline >=20 and Percentage Decrease from Baseline >=50%

Criteria 3: WOMAC Pain: decrease from baseline >=10 and Percentage Decrease from Baseline >=20%

Criteria 4: WOMAC Function: decrease from baseline >=10 and Percentage Decrease from Baseline >=20%

Criteria 5: Global Assessment: decrease from baseline >=10 and Percentage Decrease from Baseline >=20%

A subject is a 'Yes' responder if either of criteria 1 or 2 are satisfied. If neither criteria 1 or 2 are satisfied, criteria 3, 4 and 5 will be

checked. A subject is a 'Yes' responder if at least 2 of these 3 criteria (3, 4, 5) are satisfied.

Programming notes: Criteria column will be flagged with the number 1, 2, 3, 4, 5 only if the conditions for that criteria are satisfied.

Criteria 3, 4, 5 will be shown only if Crteria 1 and 2 have been checked and neither of these intial two conditions are satisfied.

Final 1.0

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Listing 16.2.6.20 Global Improvements

Treatment = MIV-711 200 mg

Date

Of Patient Visit Assessment

Knee problem

Knee Pain

Knee Function

Medivir

Final 1.0 Protocol: MIV-711-201 22 June 2017

Medivir

Protocol Number: MIV-711-201

Listing 16.2.6.21 Quality of Life Patient Reported Outcomes - EQ-5D-5L

Treatment = MIV-711 200 mg

Date

Of Usual Pain or Anxiety or Health rating Visit Assessment Mobility Self-care activity Discomfort depression Patient score

Page X of Y

Medivir
Protocol: MIV-711-201
22 June 2017

Protocol Number: MIV-711-201

Listing 16.2.6.22

Quality of Life Patient Reported Outcomes Change from Baseline Scores - EQ-5D-5L

Treatment = MIV-711 200 mg

Date
Of Usual Pain or Anxiety or Health rating
Patient Visit Assessment Mobility Self-care activity Discomfort depression score

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Listing 16.2.6.23
Brief Medication Questionnaire

Treatment = MIV-711 200 mg

Date Of

Patient Visit Assessment

Question

Response

How much did you take each time How many days did you take it The dosage times are inconvenient Etc...

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Listing 16.2.6.24 E-Diary Assessments over the Last 12 Hours

Treatment = MIV-711 200 mg

Pain NRS: Overall medication pain severity use over in target Date last 12 Pain medication usage knee over Of Patient Visit Assessment hours? over last 12 hours last 12 hours IMP Intake

YES Less than Normal NO Normal

More than normal


Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Listing 16.2.6.25
Efficacy Biomarkers from Serum and Urine Samples

Treatment = MIV-711 200 mg

Patient

Date

Of

Visit Assessment CTX-I

II II

urine CTX-

Serum


Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Listing 16.2.6.26
Time-Integrated Concentrations (TIC) and Their Z-scores for Efficacy Biomarkers from Serum and Urine Samples

Treatment = MIV-711 200 mg

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Listing 16.2.7.1 Adverse Events

| | Adverse Event<br>>MedDRA Preferred Term | Start<br>Date | Stop<br>Date | Seri- | | | Action<br>Taken<br>Study<br>Medica-<br>tion | Relation-<br>ship to<br>Study<br>Medica- | AE<br>Start<br>Time<br>from<br>First<br>Dose |
|---|---|---|---|---|---|---|---|---|---|
| Patient | >>System Organ Class | Time | Time | ous | Outcome | Severity | [1] | tion | (day) |

<sup>[1]</sup> Action taken results that state 'MEDICATION' indicate a concomitant medication was administered. No action was taken with respect to study medication unless specifically stated otherwise

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Listing 16.2.7.2 Serious Adverse Events

| | | | | | | | | AE |
|---|---|---|---|---|---|---|---|---|
| | | | | | | Action | | Start |
| | | | | | | Taken | Relation- | Time |
| | | | | | | Study | ship to | from |
| | Adverse Event | Start | Stop | | | Medica- | Study | First |
| | >MedDRA Preferred Term | Date | Date | | | tion | Medica- | Dose |
| Patient | >>System Organ Class | Time | Time | Outcome | Severity | [1] | tion | (day) |

<sup>[1]</sup> Action taken results that state 'MEDICATION' indicate a concomitant medication was administered. No action was taken with respect to study medication unless specifically stated otherwise

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Listing 16.2.7.3
Adverse Events Leading To Discontinuation

| | | | | | | | Action<br>Taken | Relation- | AE<br>Start<br>Time |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | Study | ship to | from |
| | Adverse Event | Start | Stop | | | | Medica- | Study | First |
| | >MedDRA Preferred Term | Date | Date | Seri- | | | tion | Medica- | Dose |
| Patient | >>System Organ Class | Time | Time | ous | Outcome | Severity | [1] | tion | (day) |

<sup>[1]</sup> Action taken results that state 'MEDICATION' indicate a concomitant medication was administered. No action was taken with respect to study medication unless specifically stated otherwise

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Listing 16.2.8.1 Clinical Laboratory Chemistry - Observed Values

Treatment = MIV-711 200 mg

| | | | | Lab | Lab | Lab | Lab |
|---|---|---|---|---|---|---|---|
| | | Collection | Collection | Parameter 1 | parameter 2 | parameter 3 | parameter 4 |
| Patient | Visit | Date | Time | (unit) | (unit) | (unit) | (unit) |
| | | | | Result/Flag | Result/Flag | Result/Flag | Result/Flag |

H=High, L=Low, CS=Clinically Significant, NCS=Not Clinically Significant

Programming Note: If Flag is present (H or L), clinical significance will be identified by one of 'NCS' or 'CS'.

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Listing 16.2.8.2 Clinical Laboratory Hematology - Observed Values

Treatment = MIV-711 200 mg

| | | | | Lab | Lab | Lab | Lab |
|---|---|---|---|---|---|---|---|
| | | Collection | Collection | Parameter 1 | parameter 2 | parameter 3 | parameter 4 |
| Patient | Visit | Date | Time | (unit) | (unit) | (unit) | (unit) |
| | | | | Result/Flag | Result/Flag | Result/Flag | Result/Flag |

H=High, L=Low, CS=Clinically Significant, NCS=Not Clinically Significant

Programming Note: If Flag is present (H or L), clinical significance will be identified by one of 'NCS' or 'CS'.

Medivir

Final 1.0 Protocol: MIV-711-201 22 June 2017

Medivir Page X of Y

Protocol Number: MIV-711-201

Listing 16.2.8.3 Clinical Laboratory Urinalysis - Observed Values

Treatment = MIV-711 200 mg

| | | | | Lab | Lab | Lab | Lab |
|---|---|---|---|---|---|---|---|
| | | Collection | Collection | Parameter 1 | parameter 2 | parameter 3 | parameter 4 |
| Patient | Visit | Date | Time | (unit) | (unit) | (unit) | (unit) |
| | | | | Result/Flag | Result/Flag | Result/Flag | Result/Flag |

H=High, L=Low, AB=Abnormal, CS=Clinically Significant, NCS=Not Clinically Significant

Programming Note: If Flag is present (H, L, or AB), clinical significance will be identified by one of 'NCS' or 'CS'.

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Listing 16.2.8.4

Clinical Laboratory Urinalysis - Positive Microscopic Findings

Treatment = MIV-711 200 mg

| | | Collection | Collection | | | | | Clinical |
|---|---|---|---|---|---|---|---|---|
| Patient | Visit | Date | Time | Test Name | Result | Unit | Flag | Significance |

\*H=High, L=Low, AB=Abnormal, CS=Clinically Significant, NCS=Not Clinically Significant

Programming Note: If Flag is present (H, L, or AB), clinical significance will be identified by one of 'NCS' or 'CS'.

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Listing 16.2.8.5
Vital Signs - Observed Values

| | | | | Supine | Supine<br>Systolic<br>Blood | Supine<br>Diastolic<br>Blood | Pulse | Body |
|---|---|---|---|---|---|---|---|---|
| Patient | Visit | Collection<br>Date | Collection<br>Time | Heart Rate (beats/min) | Pressure<br>(mmHg) | Pressure<br>(mmHg) | Oximetry<br>(%) | Temperature (°C) |

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Listing 16.2.8.6
Vital Signs Change from Baseline

| | | | | Supine | Supine<br>Systolic<br>Blood | Supine<br>Diastolic<br>Blood |
|---|---|---|---|---|---|---|
| Patient | Visit | Collection<br>Date | Collection<br>Time | Heart Rate (beats/min) | Pressure<br>(mmHg) | Pressure<br>(mmHg) |

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Listing 16.2.8.7

Vital Signs Overall Qualitative Results Abnormal Assessments

Treatment = MIV-711 200 mg

Collection Collection

Patient Visit Date Time Assessment Interpretation

ABNORMAL, NCS ABNORMAL, CS

NCS = Not Clinically Significant, CS = Clinically Significant

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Listing 16.2.8.8
12 Lead ECG Quantitative Findings

Treatment = MIV-711 200 mg

| | | | 0.11 | 0.11 | Heart | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Collect- | Collec- | Rate | | | 27.2 | 0.00 | | |
| | | | ion | tion | (beats | PR | RR | QRS | QΤ | QTcB | QTcF |
| Patient | Visit | Timepoint | Date | Time | /min) | (msec) | (msec) | (msec) | (msec) | (msec) | (msec) |

QTCB = QT corrected according to Bazett, QTCF = QT corrected according to Fridericia.

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Listing 16.2.8.9
12 Lead ECG Change From Baseline

Treatment = MIV-711 200 mg

| | | | Collection | Collection | QT | QTcB | QTcF |
|---|---|---|---|---|---|---|---|
| Patient | Visit | Timepoint | Date | Time | (msec) | (msec) | (msec) |

 ${\tt QTcB} = {\tt QT}$  corrected according to Bazett,  ${\tt QTcF} = {\tt QT}$  corrected according to Fridericia.

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Listing 16.2.8.10
12 Lead ECG Overall Qualitative Assessment

Treatment = MIV-711 200 mg

Collection Collection Assess-Patient Visit Timepoint Date Time ment Interpretation Comment

NCS = Not Clinically Significant, CS = Clinically Significant

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Listing 16.2.8.11
Physical Examination Abnormal Findings

Treatment = MIV-711 200 mg

Exam Exam Clinical
Patient Visit Date Time Body System Abnormality Significance

NCS

CS

NCS = Not Clinically Significant, CS = Clinically Significant

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Listing 16.2.8.12 Patient Weight

Treatment = MIV-711 200 mg

Patient Visit Date Time Weight (kg)

Medivir

Protocol: MIV-711-201

Final 1.0 22 June 2017

Medivir

Protocol Number: MIV-711-201

Page X of Y

Listing 16.2.8.13
Phone Call to Assess Safety

Treatment = MIV-711 200 mg

Patient Visit Comments